Once-Yearly Zoledronic Acid for Treatment of Postmenopausal Osteoporosis (HORIZON - Pivotal Fracture Trial, PFT)

**DUPLICATE HORIZON-PFT** 

February 11, 2021

NCT00049829

#### 1. RCT Details

This section provides a high-level overview of a **published** RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Once-Yearly Zoledronic Acid for Treatment of Postmenopausal Osteoporosis (HORIZON - Pivotal Fracture Trial, PFT)

#### 1.2 <u>Intended aim(s)</u>

To assess the effects of 15-minutes annual infusions of zoledronic acid (5mg) on hip fracture risk in postmenopausal women with osteoporosis during a 3-year period.

#### 1.3 Primary endpoint for replication

Co-primary endpoints were incidence of hip fracture and incidence of vertebral fracture. We focus on the risk of hip fracture for replication.

#### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

Assuming a 3-year fracture rate of 1.8% in the placebo group, it was determined that with 7,400 patients the log-rank test had a power of 90% (with a two-sided alpha of 0.05) to detect a 50% reduction in hip fractures.

#### 1.5 Secondary endpoint for replication (assay sensitivity) and RCT finding

Non-vertebral fracture

#### 1.6 <u>Trial estimate</u>

Hazard Ratio, HR = 0.59 (95% CI, 0.42 to 0.83) comparing zoledronic-acid group vs. placebo group during a 3-year period (Black et al., 2007).

Note. The follow-up period of the RWE replication is set at 18months. In the trial, the HR comparing zoledronic-acid group vs. placebo group during an 18-month period is estimated to be  $\sim 0.745$ . The HR at 18 months is defined as the ratio between the cumulative incidences of hip fracture events in the zoledronic-acid and placebo groups ( $HR = \frac{CI_{ZA}}{CI_{placebo}}$ ) measured after 18 months of follow-up. The estimates of the cumulative incidences of hip fracture events have been extracted by the Kaplan-Meier curves reported in the trial using a dedicated software (Graph Grabber 2.0.2, Quintessa Ldt).

#### 2. Person responsible for implementation of replication in Action

Elvira D'Andrea, MD, MPH, implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of the design and analytic choices. All implementation steps are recorded, and the implementation history is archived in the platform.

#### 3. Data Source(s)

Optum CDM, IBM® MarketScan®

#### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Cohort Entry Date (Day 1) [Dispensation of Zoledronic acid (5 mg, IV administered annually)] OR [Raloxifene (oral tablet administered daily)] INCL: Diagnosis of Osteoporosis Days [Enrollment, 0] **INCL**: Use of meds for osteoporosis <u>INCL</u>: Age ≥ 65 Days [0] EXCL: Amputation or absence of lower limb Days [Enrollment, 0] EXCL: Prior use of Bisphosphonate OR parathyroid hormon Days [-730, 0] EXCL: Treatment and Prevention of Glucocorticoid-Induced Osteoporosis Days [-730, 0] EXCL: Treatment of Paget's Disease of Bone Days [-730, 0] Days [-450, 0] EXCL: Life expectancy less than 6 months (CCl ≥ 10)

Days [-450, 0] EXCL: Malignant neoplasms Days [-365, 0] ons that influence bone metabolism (e.g frome, Anorexia, bulimia, RA, SLE, IBD, hyperthyroidism, etc.) Days [-365, 0] EXCL: conditions/circumstances likely to lead to poor treatment adherence (Alcohol/drug abuse)

Days [-365, 0] or GH Days [-180, 0] EXCL: End-Stage Liver Disease Days [-180, 0] EXCL: End-Stage Renal Disea Days [-180, 0] Days [-180, 0] EXCL: Pregnancy Days [-180, 0] EXCL: Prior use of oral corticosteroids Days [-30, 0] PRIMARY OUTCOME: Hip fractures Covariate Assessment Window Days [-450, 0] Follow Up Window Days [1, censor<sup>a</sup>] <sup>a</sup> Censoring criteria: Day 0 Occurrence of outcome Death Disenrollment Nursing home admission Specific date reached End of index exposure

Figure 1. Design Diagram - HORIZON-PFT TRIAL REPLICATION

#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing 15-minute annual infusions of zoledronic acid (5mg) to raloxifene (as a proxy for placebo). Raloxifene was selected as the placebo proxy because raloxifene was the most common concomitant osteoporosis medication used in the trial in both study arms. In addition, prior evidence indicates no effect of raloxifene on the primary outcome of hip fracture (Ettinger et al., 1999, Ensrued et al., 2008). The patients will be required to have continuous enrollment during a baseline period of 450 days (15 months) before initiation of zoledronic acid or comparator. We will restrict the analyses to women, older than 65, with osteoporosis.

#### 5.2 Important steps for cohort formation

New use of zoledronic acid (exposure) is defined as no use of the exposure drug in the 450 days prior to index date. New users of zoledronic acid will be allowed to receive concomitant therapy with raloxifene before and/or during the study period, similar to the trial. We use the long look-back period of 450 days to define new use because zoledronic acid is given as a yearly infusion; thus, a identifying whether a patient has current zoledronic acid exposure requires at least 365 days of look back. We extended this lookback to 450 days (approximately 15 months) to allow for patients who have a short gap between infusions. To keep the amount of lookback available in the 2 treatment groups equal, New use of raloxifene (comparator, proxy to placebo) was also defined as no use of either exposure or comparator drugs in the 450 days prior to index date.

#### 5.2.1 Eligible cohort entry dates

Zoledronic acid indication for treatment of postmenopausal women with osteoporosis was approved by FDA on Aug 20, 2007.

- IBM® MarketScan®: Aug 21, 2007 December 31, 2018 (end of available data)
- Optum CDM: Aug 21, 2007 Mar 31, 2020 (end of available data)

# 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

#### 5.3 Flowchart of the study cohort assembly

For zoledronic acid vs. raloxifene

| | Optı | ım CDM | IBM® Ma | rketScan® |
|---|---|---|---|---|
| | Excluded Patients | Remaining Patients | Excluded Patients | Remaining Patients |
| All patients | | 77,673,639 | | 200,203,908 |

| | -77,476,067 | 197,572 | - | 489,107 |
|---|---|---|---|---|
| Did not meet cohort entry criteria | | | 199,714,801 | |
| Excluded due to insufficient enrollment | -52,317 | 145,255 | -164,242 | 324,865 |
| Excluded due to prior use of referent | -81,791 | 63,464 | -185,458 | 139,407 |
| Excluded due to prior use of exposure | -9,268 | 54,196 | -29,153 | 110,254 |
| Excluded because patient qualified in >1 exposure category | -1 | 54,195 | -1 | 110,253 |
| Excluded based on Inclusion #1 - Age, range 65-89 years | -17,914 | 36,281 | -58,739 | 51,514 |
| Excluded based on Inclusion #2 - Gender, female [Excluded if Male or Unknown] | -6,080 | 30,201 | -6,857 | 44,657 |
| Excluded based on Inclusion #3 - Osteoporosis | -3,624 | 26,577 | -3,936 | 40,721 |
| Excluded based on Exclusion #1 - Oral bisphosphonate use | -6,854 | 19,723 | -10,259 | 30,462 |
| Excluded based on Exclusion #2.1 - PTH or PTH analogue use | -305 | 19,418 | -814 | 29,648 |
| Excluded based on Exclusion #2.2 - Anabolic–androgenic steroids (AAS) and | -10 | 19,408 | -32 | 29,616 |
| growth hormones (GH) | | | | |
| Excluded based on Exclusion #2.3 - Glucocorticoids use | -1,352 | 18,056 | -1,697 | 27,919 |
| Excluded based on Exclusion #3 - CCI (180 days) >=10 | -196 | 17,860 | -154 | 27,765 |
| Excluded based on Exclusion #4 - Malignant neoplasm, excluding non-melanoma | -2,461 | 15,399 | -4,141 | 23,624 |
| skin cancer | | | | |
| Excluded based on Exclusion #5 - Disorders that influence bone metabolism | -1,426 | 13,973 | -2,235 | 21,389 |
| Excluded based on Exclusion #6 - Glucocorticoid-Induced Osteoporosis | -4 | 13,969 | -5 | 21,384 |
| Excluded based on Exclusion #7 - Paget's Disease | -43 | 13,926 | -65 | 21,319 |
| Excluded based on Exclusion #8 - Alcohol abuse or Drug addiction or Non- | -141 | 13,785 | -137 | 21,182 |
| compliance | 1 | 10.504 | 2 | 21 170 |
| Excluded based on Exclusion #9 - Pregnancy | -1 | 13,784 | -3 | 21,179 |
| Excluded based on Exclusion #10 - Lower extremity amputation | -18 | 13,766 | -37 | 21,142 |
| Excluded based on Exclusion #11 - Denosumab use | -53 | 13,713 | -35 | 21,107 |
| Excluded based on Exclusion #12 - Zoledronic Acid use (for raloxifene users) | -223 | 13,490 | -313 | 20,794 |
| Excluded based on Exclusion criteria #13 - End-stage renal disease | -5 | 13,485 | -12 | 20,782 |
| Excluded based on Exclusion criteria #14 - End-stage liver disease | -33 | 13,452 | -66 | 20,716 |
| Excluded based on Exclusion criteria #15 - Blindness or low vision | -32 | 13,420 | -25 | 20,691 |
| Excluded based on Exclusion criteria #16 - Abaloparatide | -0 | 13,420 | -0 | 20,691 |
| Excluded based on Exclusion criteria #17 - Romosozumab | -0 | 13,420 | -0 | 20,691 |
| Final cohort | | 13,420 | | 20,691 |

#### 6. Variables

#### 6.1 Exposure-related variables:

#### Study drug:

The study exposure of interest is new initiation of zoledronic acid 5 mg, IV administered annually. New initiation will be defined by no use of zoledronic acid in the prior 15 months (450 days) before treatment initiation (washout period).

#### Comparator agents:

#### Primary analysis:

- New initiators of raloxifene, oral tablet administered daily. New initiation will be defined by no use of raloxifene and zoledronic acid in the prior 15 months (450 days) before treatment initiation (washout period).

#### Secondary analysis:

- Non-user comparator (risk-set sampled cohort).

#### 6.2 Preliminary Covariates:

- Age
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date.

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (**Appendix B**). Gender is not included since the study is already restricted to female subjects.

#### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcome variables of interest (definitions provided in **Appendix A**):

Primary outcome: Hip fracture

- Secondary outcome:
  - o Non-vertebral fracture

#### 6.3.2 Study follow-up

Intention-to-treat (ITT) analysis will be conducted with treatment defined as the index drug on day of cohort entry. Because the exposure (zoledronic acid) is administered annually, patients receiving the exposure are automatically covered with medication for at least 12 months. In addition, the comparator (raloxifene) is intended to proxy for placebo, so nonadherence to the comparator does not result in meaningful exposure misclassification. Therefore, the ITT analysis with a follow-up of 18 months (540 days) will be the primary analysis.

The follow-up will start the day after drug initiation (i.e., cohort entry date), as described in the HORIZON-PFT, and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a
    patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same
    reason.

#### 7. Initial Feasibility Analysis

#### Action report name:

For zoledronic acid vs. raloxifene

Optum CDM- <a href="https://bwh-dope.aetion.com/projects/details/1406/results/60058/result/0">https://bwh-dope.aetion.com/projects/details/1406/results/60058/result/0</a> IBM® MarketScan®- <a href="https://bwh-dope.aetion.com/projects/details/1407/results/60060/result/0">https://bwh-dope.aetion.com/projects/details/1406/results/60058/result/0</a>

Date conducted: 10/17/2020

Complete Action feasibility analysis using age and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

• Report patient characteristics by treatment group

### • For zoledronic acid vs. raloxifene

| | | Optum CDM | | IBM® MarketScan® | | |
|---|---|---|---|---|---|---|
| Variable | Raloxifene -<br>Comparator | Zoledronic Acid -<br>Exposure | Difference | Raloxifene -<br>Reference | Zoledronic acid -<br>Exposure | Difference |
| Number of patients | 6,815 | 6,605 | - | 6,694 | 13,997 | - |
| Age | | | | | | |
| mean (sd) | 73.41 (5.90) | 74.02 (5.52) | -0.62 (-0.81, -<br>0.42) | 73.81 (7.06) | 75.61 (7.14) | -1.80 (-2.01, -<br>1.60) |
| median [IQR] | 73.00 [68.00,<br>78.00] | 75.00 [69.00,<br>79.00] | - | 72.00 [68.00,<br>79.00] | 75.00 [70.00,<br>81.00] | - |
| Combined<br>Comorbidity Score -<br>CCI (180 days) | | | | | | |
| mean (sd) | 1.38 (1.52) | 1.49 (1.56) | -0.11 (-0.16, -<br>0.06) | 0.96 (1.20) | 1.22 (1.35) | -0.27 (-0.30, -<br>0.23) |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | - |

- Report summary parameters of study population FEASIBILITY- FOR STUDY OUTCOME
   For zoledronic acid vs. raloxifene

| | Optum CDM | IBM®<br>MarketScan® |
|---|---|---|
| Number of patients in full cohort | 13,420 | 20,691 |
| Number of patients dropped as incomplete cases | 0 | 0 |
| Number of patients that did not begin follow-up | 0 | 0 |
| Number of patients in analytic cohort | 13,420 | 20,691 |
| Number of events | 146 | 208 |
| Number of person-years | 16,243 | 24,519 |
| Number of patients in group: Raloxifene - Comparator | 6,815 | 6,694 |
| Number of patients in group: Zoledronic Acid - Exposure | 6,605 | 13,997 |
| Risk per 1,000 patients | 10.88 | 10.05 |
| Rate per 1,000 person-years | - | - |

- Report median follow-up time by treatment group
   For zoledronic acid vs. raloxifene

| Median Follow-Up Time (Days) [IQR] – ITT analysis | | |
|---|---|---|
| Patient Group Optum CDM IBM® MarketScan® | | |
| Overall Patient Population | 540 [375, 540] | 540 [340, 540] |
| Referent - Raloxifene | 540 [363, 540] | 540 [363, 540] |
| Exposure - ZA | 540 [383, 540] | 540 [329, 540] |

- Report reasons for censoring in the overall study population
   For zoledronic acid vs. raloxifene

| Reasons | Optum CDM | IBM®<br>MarketScan® |
|---------------------------|---------------|---------------------|
| Overall | 10750 | 17260 |
| Outcome | 146 (1.1%) | 208 (1.0%) |
| Death | 0 (0.0%) | 62 (0.3%) |
| Maximum follow-up time | 8,891 (66.3%) | 13,112 (63.4%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 2,589 (19.3%) | 5,969 (28.8%) |
| Nursing home Occurred | 838 (6.2%) | 630 (3.0%) |

• Report overall risk of the primary outcome.

| | Optum CDM | IBM®<br>MarketScan® | Pooled |
|-------------------------|-----------|---------------------|--------|
| Risk per 1,000 patients | 10.9 | 10.1 | 10.4 |

#### 8. Initial Power Assessment

### Action report name:

For zoledronic acid vs. raloxifene

Optum CDM- https://bwh-dope.aetion.com/projects/details/1406/results/60059/result/0

IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1407/results/60061/result/0

Date conducted: 10/17/2020

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 2 covariates: age and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

• Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.

#### o Pooled

| o <u>Pooled</u> | 1 |
|----------------------------|-------------|
| Superiority Analysis | |
| Number of patients matched | 25,518 |
| Reference | 12,759 |
| Exposed | 12,759 |
| Risk per 1,000 patients | 10.40 |
| Desired HR from RCT | 0.59 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 265.3872 |
| Power | 0.990300973 |

o Optum CDM

| Companie vite Amelouie | |
|----------------------------|-------------|
| Superiority Analysis | |
| Number of patients matched | 12,130 |
| Reference | 6,065 |
| Exposed | 6,065 |
| Risk per 1,000 patients | 10.90 |
| Desired HR from RCT | 0.59 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 132.217 |
| Power | 0.858487133 |

### o <u>IBM® MarketScan®</u>

| Superiority Analysis | |
|----------------------------|------------|
| Number of patients matched | 13,388 |
| Reference | 6,694 |
| Exposed | 6,694 |
| Risk per 1,000 patients | 10.10 |
| Desired HR from RCT | 0.59 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 135.2188 |
| Power | 0.86602361 |

• Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 10/29/20 |
|-------------------------|------------------|----------------|----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 11/15/20 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

#### Action report name:

For zoledronic acid vs. raloxifene

Optum CDM: https://bwh-dope.aetion.com/projects/details/1406/results/64560/result/0

IBM® MarketScan®: https://bwh-dope.aetion.com/projects/details/1407/results/64559/result/0

Date conducted: 01/19/2021

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to **Appendix B**.

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---------------------------|----------------|---------------|---------------|
| Dummy outcome | 697 (3.87%) | 350 (3.88%) | 347 (3.85%) |
| Death | 89 (0.49%) | 36 (0.40%) | 53 (0.59%) |
| End of index exposure | 762 (4.23%) | 372 (4.13%) | 390 (4.33%) |
| Maximum follow-up time | 11993 (66.52%) | 6058 (67.21%) | 5935 (65.84%) |
| End of patient enrollment | 4487 (24.89%) | 2198 (24.38%) | 2289 (25.39%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] – ITT analysis | | |
|---|---|---|
| Patient Group Optum CDM IBM® MarketScan® | | |
| Overall Patient Population | 540 [404.5, 540] | 540 [365, 540] |
| Referent - Raloxifene | 540 [426, 540] | 540 [365, 540] |
| Exposure - ZA | 540 [386, 540] | 540 [364.5, 540] |

• Report overall risk of the primary outcome.

| | Optum CDM | IBM® MarketScan® | Pooled |
|-------------------------|-----------|------------------|--------|
| Risk per 1,000 patients | 10.9 | 10.1 | 10.4 |

#### 10. Final Power Assessment

Date conducted: 01/19/2021

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

# o <u>Pooled</u>

| 18,028 |
|-------------|
| 9,014 |
| 9,014 |
| 10.40 |
| 0.59 |
| 0.05 |
| 187.4912 |
| 0.950774073 |

### o Optum CDM

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 6,396 |
| Reference | 3,198 |
| Exposed | 3,198 |
| Risk per 1,000 patients | 10.90 |
| Desired HR from RCT | 0.59 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 69.7164 |
| Power | 0.595938014 |

o IBM® MarketScan®

| O IBIVIO IVIGINOUS CALLO | |
|----------------------------|-------------|
| Superiority Analysis | |
| Number of patients matched | 11,632 |
| Reference | 5,816 |
| Exposed | 5,816 |
| Risk per 1,000 patients | 10.10 |
| Desired HR from RCT | 0.59 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 117.4832 |
| Power | 0.815816276 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 01/19/21 |
|-------------------------|------------------|----------------|----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 01/19/21 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 11. Study Confidence and Concerns

<u>Deadline for voting on study confidence and listing concerns:</u>

Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the success of the RWD study in the Google Form. This form also provides space for reviewers to list any concerns that they feel may contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study variables, or residual confounding.

All responses will be kept confidential and individual-level results will only be shared with the individual respondent.

• After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

#### 12. Register study protocol on clinicalTrials.gov

#### Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

#### 13. Comparative Analyses

#### Action report name:

Date conducted:

#### 13.1 For primary analysis:

In the PS-matched cohort from Section 9, to estimate the risk of hip fracture for zoledronic acid users versus raloxifene users during an 18-month period using a Cox regression hazard regression model.

#### 13.2For sensitivity analyses:

#### **Secondary analyses:**

- In the PS-matched cohort from Section 9, to estimate the risk of non-vertebral fracture for zoledronic acid users versus raloxifene users during an 18-month period using a Cox regression hazard regression model.
- To estimate the risk of hip fracture for zoledronic acid versus non-user comparator using a risk-set sampled cohort.

<u>Subgroup analysis</u>: In the PS-matched cohort from Section 9, to estimate the risk of hip fracture stratified by age (women younger or older than 75 years). The estimates are compared with the results from a post-hoc analysis of the Horizon-PFT on women older than or equal to 75 (Boonen et al.).

### 14. Requested Results

### 14.1 Table 1: Baseline characteristics before and after adjustment

| Variable | 9, | After adjustment | | | |
|--------------------|----|------------------|----------|------------|---|
| | | Referent | Exposure | Std. diff. | |
| Number of patients | | - | | | - |
| Age categories | | | | | |
| ••• | | | | | |

### 14.2 Table 2: Follow-up time

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

### 14.3 Table 3: Censoring events

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

#### 14.4 Table 4: Results from primary analysis

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

#### 14.5 Table 5: Results from secondary analyses

#### 15. References

Black DM, Delmas PD, Eastell R, Reid IR, Boonen S, Cauley JA, Cosman F, Lakatos P, Leung PC, Man Z, Mautalen C, Mesenbrink P, Hu H, Caminis J, Tong K, Rosario-Jansen T, Krasnow J, Hue TF, Sellmeyer D, Eriksen EF, Cummings SR; HORIZON Pivotal Fracture Trial. Once-yearly zoledronic acid for treatment of postmenopausal osteoporosis. N Engl J Med. 2007 May 3;356(18):1809-22. doi: 10.1056/NEJMoa067312.

Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

Ensrud KE, Stock JL, Barrett-Connor E, Grady D, Mosca L, Khaw KT, Zhao Q, Agnusdei D, Cauley JA. Effects of raloxifene on fracture risk in postmenopausal women: the Raloxifene Use for the Heart Trial. Journal of bone and mineral research. 2008 Jan;23(1):112-20.

Ettinger B, Black DM, Mitlak BH, Knickerbocker RK, Nickelsen T, Genant HK, Christiansen C, Delmas PD, Zanchetta JR, Stakkestad J, Glüer CC. Reduction of vertebral fracture risk in postmenopausal women with osteoporosis treated with raloxifene: results from a 3-year randomized clinical trial. Jama. 1999 Aug 18;282(7):637-45.

Wright NC, Daigle SG, Melton ME, Delzell ES, Balasubramanian A, Curtis JR. The Design and Validation of a New Algorithm to Identify Incident Fractures in Administrative Claims Data. J Bone Miner Res. 2019 Oct;34(10):1798-1807. doi: 10.1002/jbmr.3807.

Boonen S, Black DM, Colón-Emeric CS, et al. Efficacy and safety of a once-yearly intravenous zoledronic acid 5 mg for fracture prevention in elderly postmenopausal women with osteoporosis aged 75 and older. J Am Geriatr Soc. 2010;58(2):292-299. doi:10.1111/j.1532-5415.2009.02673.x

| # | HORIZON-PFT trial definitions | Implementation in routine care | Please see the following Googl<br>https://drive.google.com/drive/folde | ogle Drive for further details or any missing information: olders/1WD618wrywYjEaXzfl_TcuK-VCcnb6b-gV?usp=sharing |
|---|---|---|---|---|
| | Trial details - clinicaltrial.gov NCT00049829 | | 10 code lists will be available in the above Google E<br>using a SAS macro that implements forwar | of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-<br>prive Folder (link above). ICD-9 to ICD-10 code conversions were completed<br>d/ backward mapping based on the CMS ICD-9 to ICD-10 mapping:<br>10-cm-and-nex-crosswalk-general-equivalence-mapping.html |
| | EXPOSURE vs. | COMPARISON | References/Rationale | Color coding |
| | Exposure: Zoledronic acid (5 mg) 15-minute intravenous administration every year for 3 years vs. placebo Reference: Placebo Aim: To evaluate the effect of annual infusions of zoledronic acid on fracture risk during a 3-year period in postmenopausal women with osteoporosis All patients received oral daily calcium (1000 to 1500 mg) and vitamin D (400 to 1200 IU). | Exposure: new-use of Zoledronic acid (washout 450 days) NDC Generic Name: ZOLEDRONIC ACID ZOLEDRONIC ACID IN MANNITOL & WATER FOR INJECTION ZOLEDRONIC ACID IN MANNITOL AND 0.9 % SODIUM CHLORIDE ZOLEDRONIC ACID IN MANNITOL AND WATER FOR INJECTION ZOLEDRONIC ACID IN MANNITOL AND WATER FOR INJECTION NDC codes: 143964201, 16729024231, 17478032705, 25021080167, 42023015101, 43598033011, 47335003540, 47333096241, 54288010001, 5511106850755150026605, 67457039054, 68001036625, 78035084, 78038725, 409421501, 409421505, 16714081501, 17478032745, 23155017031, 25021080166, 45963044055, 51991006598, 53150087101, 60505611000, 63232096198, 68001036622, 78043561, 78059061, 409422801, 43598033111, 51991006498, 55111068852, 63323096600, 67457061910, 67457079410, 70860021051 CPT/HCPCS Procedure Codes: C9115, 13487, 13488, 13489, Q2051, Q4095 Reference of primary analysis: Raloxifene (proxy of placebo) Reference of primary analysis: Raloxifene (proxy of placebo) | | Criteria |
| | PRIMARY | DUTCOME | | Adequate mapping in claims |
| | Hip fracture (Dual-energy x-ray absorptiometry of the hip was performed at baseline and at months 6, 12, 24, and 36 for bone loss) - both patients in stratum 1 and stratum 2 | Measured 1 day after drug initiation (codes reported in "Hip and femur fractures codes": Hip and femur fractures Algorithm include the following case-qualifying (CO): CQ = 1 Inpatient claim with primary diagnosis code AND CQ = 2 Inpatient claim with secondary diagnosis code AND CQ = 3 Non-inpatient claim with diagnosis code AND HCPCS in (27125, 27130, 27220, 27222, 27226-27228, 27230-27248, 27254, 27254, 27267-27269, 27500-27514) OR Non-inpatient claim with diagnosis code AND ICD-9 Procedure Code in (7855, 7905, 7915, 7925, 7935, 7965, 8151, 8152) | Wright NC, Daigle SG, Melton ME, Delzell ES, Balasubramanian A, Curtis JR. The Design and Validation of a New Algorithm to Identify Incident Fractures in Administrative Claims Data J. Bone Miner Res. 2019 Oct;34(10):1798-1807. doi: 10.1002/jbmr.3807. Epub 2019 Aug S. PMID: 31170317. | Intermediate mapping in claims |
| | New Vertebral Fractures [only in patients who were not taking any osteoporosis medications at the time of randomization] only patients in stratum 1 (Spinal lateral radiographs were obtained at baseline and at 12, 24, and 36 months or early termination for patients in stratum 1 and at baseline and at 36 months or early termination for patients in stratum 2) | Measured 1 day after drug initiation: Vertebral Fractures: Algorithm include the following case-qualifying (CO): CQ = 1 Inpatient claim with primary diagnosis code AND CQ = 2 Non-inpatient claim with diagnosis code AND HCPCS in (22305, 22310, 22315, 22318, 22319, 22325-22328, 22510-22515, 22520-22525, 27200, 27202, 72291, 72292, 76012, 76013, 77082, 77085, 77086, 52360-52363) AND CQ = 3 Non-inpatient claim with diagnosis code AND HCPCS in (99024, 99058, 99201-99215, 99241-99245, 99271-99285, 99301-99355, 99366, 99385-99387,99395-99404, 99429, 99499) [Physician E&M codes] plus, up to 10 days earlier (or on the same day), Outpatient claim with HCPCS in (72010-72159, 72240-72285, 72295) [Spine imaging codes] | Outcome not included in the final analysis Wright NC, Daigle SG, Melton ME, Delzell ES, Balasubramanian A, Curtis JR. The Design and Validation of a New Algorithm to Identify Incident Fractures in Administrative Claims Data. J Bone Miner Res. 2019 Oct;34(10):1798-1807. doi: 10.1002/jbmr.3807. Epub 2019 Aug 5. PMID: 31170317. | Poor mapping or cannot be measured in claims |
| | INCLUSION | CRITERIA | | Can't be measured in claims but not important for the analysis |
| 1 | Postmenopausal women between the ages of 65 and 89 years | Female, 65-89 years at the time of drug initiation | | |
| 2 | Bone mineral density T score of -2.5 or less at the femoral neck, with or without evidence of existing vertebral fracture, or a T score of -1.5 or less, with radiologic evidence of at least two mild vertebral fractures or one moderate vertebral fracture. | Measured time of enrollment to prior to the day of drug initiation inpatient (any position), outpatient (any position): Osteoporosis diagnosis ICD-9 diagnosis: 733.00, 733.01, 733.02, 733.03, 733.09, 733.13 ICD-10 diagnosis: M81.0, M81.6, M81.8, M80.88*, M80.08* OR Measured time of enrollment to 730 days (2 years) prior to the day of drug initiation: Alendronate, Ibandronate, Risedronate, Pamidronate, Etidronate, Tiludronate | | Adequate mapping in claims of criteria extracted from clinicaltrial.gov (ESLD and Svere eye disease), after clinical review with FDA (Abaloparatide, Romosozumab) or from the protocol of Horizon-recurrent (all other criteria in blue): "Colôn-Emeric CS, Caminis J, Suh TT, Pieper CF, Janning C, Magaziner J, Adachi J, Rosario-Jansen T, Mesenbrink P, Horowitz ZD, Lyles KW; HORIZON Recurrent Fracture Trial. The PHORIZON Recurrent Fracture Trial: the prevention of subsequent fractures after low trauma hip fracture repair. Curr Med Res Opin. 2004 Jun;20(6):903-10. doi: 10.1185/03079904125003683. PMID: 15200749." Protocol of Horizon-pivotal not available - numerous unsuccessful attempts had been made to retrive it from the authors |

| | EXCLUSION | CRITERIA | |
|---|---|---|---|
| 1 | Bisphosphonate users such as Aredia® (pamidronate), Didronel® (etidronate), Fosamax® (alendronate), Actonel® (risedronate), Skelid® (tiludronate) | Measured 730 days (2 years) prior to the day of drug initiation: Generic names: Alendronate, Ibandronate, Risedronate, Pamidronate, Etidronate, Tiludronate | |
| 2.1 | Previous use of: (1) any previous use of parathyroid hormone | Measured 730 days (2 years) prior to the day of drug initiation: Generic names: Brand names: Natpara® (parathyroid hormone), Forteo®, Bonsity (teriparatide), Tymlos® (abaloparatide) | |
| 2.2 | (2) use of anabolic steroids or growth hormone within 6 months before trial entry | Measured 180 days prior to the day of drug initiation: AASs: Generic names: TESTOSTERONE, DIHYDROTESTOSTERONE PROPIONATE, ESTROGENS, ESTERIFED/METHYLTESTOSTERONE, TESTOSTERONE CYPIONATE, MICRONIZED, TESTOSTERONE CYPIONATE ESTERADIOL CYPIONATE, TESTOSTERONE ENANTHATE-ESTRADIOL OVALERATE, TESTOSTERONE MICRONIZED, TESTOSTERONE UNDEC ANOATE, METHYLTESTOSTERONE, MICRONIZED, STANOLONE, OXYMETHOLONE, NANDROLONE PIENPROPIONATE, OXANDROLONE, STANOZOLO, FLUDXYMESTERONE, TESTOSTERONE ENANTHATE, TESTOSTERONE PROPIONATE, NANDROLONE DECANOATE, METHYLTESTOSTERONE, TESTOSTERONE CYPIONATE GHS: Generic names: SOMATROPIN, TESAMORELIN ACETATE Brand names: OMNITROPE, SAIZEN, ZOMACTON, GEREF, HUMATROPE, NUTROPIN, SEROSTIM, ZORBTIVE, EGRIFTA, MACRILEN, NORDITROPIN FLEXPRO, GENOTROPIN, TEVEROPIN | |
| 2.3 | OR (3) oral or intravenous systemic corticosteroids within 12 months, | Measured 30 days prior to the day of drug initiation: Injectable (IV) or (IM): NDC Generic Name: methylprednisolone, hydrocortisone, dexamethasone CPT/HCPCS Procedure Code: J1020, J1030, J1040, J1720, J2920, J2930 Oral: NDC Generic Name: Cortisone, hydrocortisone, prednisone, prednisolone, methylprednisolone, dexamethasone CPT/HCPCS Procedure Code: J7506, J7509, J7510, J8540 | |
| 2.4 | OR (4) any previous use of strontium, or sodium fluoride within 6 months before trial entry | CRITERIA NOT APPLIED | Strontium not approved in USA for treatment of osteoprosis. Sodium Fluoride is not used to treat the osteoporosis since 2001/2002 when a RCT and sub meta-analysis showed an increased of risk of fractures in the exp |
| NA | Patients with a serum calcium level of more than 2.75 mmol per liter or less than 2.00 mmol per liter | N/A | |
| NA | Patients with a calculated creatinine clearance of less than 30.0 ml per minute at either of two baseline visits or urine dipstick results of more than 2+ for protein, without evidence of contamination or bacteriuria. | N/A | |
| NA | Written informed consent | N/A | |
| 3 | Serious disease that may limit life expectancy to less than 6 months (including sever liver and renal diseases) | Measured 180 days prior to the day of drug initiation: CCI >=10 (life expectancy less than the expected duration of the trial) | |
| 4 | New diagnosis or active treatment for any nonskin malignancy ≤ 12 months prior to randomization and any metastatic cancer | Measured 365 days prior to the day of drug initiation inpatient (any position), outpatient (any position): Malignant neoplasm; ICD-9 diagnosis: 140.xx-208.xx (except 173.xx, non-melanoma skin cancer) ICD-10 diagnosis: C00-C43, C45-C97, D45 | |

| _ | | | Measured 505 days prior to the day of drug initiation: | |
|---|---|---|---|---|
| | 5 1 | Conditions that influence bone metabolism | Anorexia and Bulimia: ICD-9 diagnosis: 307.1, 307.5x, 783.0, 783.2x,783.3,783.6,783.9 ICD-10 diagnosis: F50.xx, R63.x Cushing syndrome and disorders of adrenal glands: ICD-9 diagnosis: 255.xx ICD-10 diagnosis: E24.x Hypernarathyroidism and hyperthyroidism: ICD-9 diagnosis: 252.x ICD-10 diagnosis: 252.x Inflammatory conditions: Rheumatoid arthritis ICD-9 diagnosis: 714.0-714.4 ICD-10 diagnosis: 714.0-714.4 ICD-10 diagnosis: 715.x,M05.85x,M05.60,M08.00,M08.40 Lupus ICD-9 diagnosis: 710.0 ICD-10 diagnosis: M32.10 Crobn's disease and other IBD ICD-9 diagnosis: M32.10 Crobn's disease and other IBD ICD-9 diagnosis: S55.x, S56.x ICD-10 diagnosis: K50.xx, K51.xx | |
| | 6 | Treatment and Prevention of Glucocorticoid-Induced Osteoporosis NB. The recommended regimen is a 5 mg infusion once a year given intravenously over no less than 15 minutes. | Measured 730 days (2 years) prior to the day of drug initiation: ICD-9 diagnosis: E858.0, 962.0 Poisoning by adrenal cortical steroids, ICD-10 diagnosis: T38.0xx Adverse effect of glucocorticoids and synthetic analogues | |
| | 7 | Treatment of Paget's Disease of Bone NB. The recommended dose is a 5 mg infusion. The infusion time must not be less than 15 minutes given over a constant infusion rate. | Measured 730 days (2 years) prior to drug initiation: ICD-9 diagnosis: 731.0 Osteitis deformans without mention of bone tumor (Paget's Disease) ICD-10 diagnosis: M88.xxx Osteitis deformans [Paget's disease of bone] | |
| | 8 | Other conditions/circumstances likely to lead to poor treatment adherence | Measured 365 days prior to drug initiation in any diagnosis position in inpatient or outpatient care setting: Alcohol Abuse or Dependence ICD-9 diagnosis: 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x (CMS has not released mapping for new ICD10 for this code), V11.3x ICD-10 diagnosis: F10.x, K70.x, G62.1, I42.6, 099.31x OR Drug Abuse or Dependence ICD-9 diagnosis: 292.xx, 304.xx, 305.2x-305.9x, 648.3x ICD-10 diagnosis: F11.x, F12.x, F13.x, F14.x, F15.x, F16.x, F17.2x, F18.x, F19.x, F55.2, G62.0, 099.32x OR Non-compliance: ICD-9 diagnosis: V45.12, V15.81 ICD-10 diagnosis: Z91.19, Z91.15 | |
| | 9 | Pregnancy (even though it is very unlikely to found cases we add this criteria to make sure all women are postmenopausal) | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting Pregnancy (see "Pregnancy codes") | |
| 1 | | Low fracture risk or unlikely to benefit:<br>Amputee | Measured time of enrollment to prior to the day of drug initiation inpatient (any position), outpatient (any position): ICD-9 Diagnosis: Acquired absence of lower limb: V49.7x, Traumatic amputation 895.x, 896.x, 897.x ICD-9 Procedure: Amputation Of Lower Limb: 84.1xx, 84.25-84.28 ICD-10 Diagnosis: Acquired absence of lower limb: Z89.4xx, Z89.5xx, Z89.6xx, Traumatic amputation: S78.xxx ICD-10 Procedure: Detachment of lower limb: 0Y6xxx | |
| 1 | 11 | Zoledronic acid use (to exclude ZA use in the raloxifene group) | Measured 450 (I year + 90 days) prior to the day of drug initiation:<br>(same as exposure) | |
| 1 | 12 | Denosumab use | Measured 450 (1 year +90 days) prior to the day of drug initiation: | |
| | | | | 1 |

| 13 | End-Stage Renal Disease | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: 2 codes for occurrence of ESRD/dialysis (either inpatient or outpatient), separated by at least 30 days: ICD-9 Diagnosis: S85.6, V45.1, V56.0, V56.8, 585.5 ICD-9 Procedure: 39.95, 54.98 ICD-10 Diagnosis: N18.5, N18.6, Z49.31, Z49.32, Z99.2 ICD-10 Procedure: 39.95, 54.98 ICD-10 Procedure: 3EIM392, SA1D60Z, SA1D00Z, 3EIM39Z, SA1D60Z, 5A1D00Z ICD-10 Procedure: 3EIM39Z, SA1D60Z, 5A1D00Z, 3EIM39Z, SA1D60Z, 5A1D00Z ICD-10 Procedure: 3EIM39Z, SA1D60Z, S01D00Z, 3EIM39Z, SA1D60Z, 5A1D00Z ICD-10 Procedure: 3EIM39Z, SA1D60Z, S01D00Z, 3EIM39Z, SA1D60Z, SA1D00Z ICD-10 Procedure: 3EIM39Z, SA1D60Z, S01D00Z, S | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagifilozian vicrus other non-giffilozian atidabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagifilozia and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagifilozia Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAH.118.039177 |
|---|---|---|---|
| | | OR <u>Kidney transplant:</u> ICD-9 Diagnosis: 996.81, V42.0 ICD-9 Procedure: 55.6, 55.69 ICD-10 Diagnosis: 786.10, T86.13, T86.19, Z48.22, Z94.0, T86.11, T86.12 ICD-10 Procedure: 0T700Z0, 0T700Z2, 0TY10Z0, 0TY00Z1, 0TY10Z1, 0TY10Z2 <u>WICDS-CPT_Code-S0366</u> , S0365 | |
| 14 | End-Stage Liver Disease | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: Cirrhosis. ICD-9 Diagnosis: 571.2, 571.5, 571.6 ICD-10 Diagnosis: K70.11, K70.2, K70.3x, K70.4x, K74.x Hepatic decompensation: ICD-9 Diagnosis: 456.0, 456.20, 456.1, 456.21, 789.5, 789.59, 572.2, 567.0, 567.2, 567.21, 567.22, 567.29, 567.8, 567.89, 567.89, 567.9, 572.4 ICD-10 Diagnosis: R18.x, 185.x, K72.x, K65.x, K66.x, K67 HCC is already excluded with exclusion criteria 4 | |
| 15 | Blindness or compromised vision | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: ICD-9 Diagnosis: 369.x ICD-10 Diagnosis: H54.x | |
| 16 | Abaloparatide | Measured 450 (1 year +90 days) prior to the day of drug initiation:<br>Generic name:<br>Abaloparatide | |
| 17 | Romosozumab | Measured 450 (1 year + 90 days) prior to the day of drug initiation:<br>Generic name:<br>Romosozumab | |

#### HIP AND FEMUR FRACTURES CODES ICD9 Diagnosis codes (excluding rare fractures in young children) Fracture of neck of femur 820 Fracture of neck of femur 820.0 Closed fracture of intracapsular section 820.00 Closed fracture of intracapsular section of neck of femur, unspecified 820.02 Closed fracture of midcervical section of neck of femur 820.03 Closed fracture of base of neck of femur 820.09 Other closed transcervical fracture of neck of femur 820.1 Open fracture of intracapsular section of neck of femur 820.10 Open fracture of intracapsular section of neck of femur, unspecified 820.11 Open fracture of epiphysis (separation) (upper) of neck of femur 820.12 Open fracture of midcervical section of neck of femur 820.13 Open fracture of base of neck of femur 820.19 Other open transcervical fracture of neck of femur 820.2 Closed fracture of trochanteric section 820,20 Closed fracture of trochanteric section of neck of femur 820.21 Closed fracture of intertrochanteric section of neck of femur 820.22 Closed fracture of subtrochanteric section of neck of femur 820.3 Open fracture of trochanteric section 820.30 Open fracture of trochanteric section of neck of femur, unspecified 820.31 Open fracture of intertrochanteric section of neck of femur 820.32 Open fracture of subtrochanteric section of neck of femur 820.8 Closed fracture of unspecified part of neck of femur 820.9 Open fracture of unspecified part of neck of femur Fracture of other and unspecified parts of femur 821 Closed fracture 821.0 Closed fracture of femur 821.00 Closed fracture of unspecified part of femur 821.01 Closed fracture of shaft of femur convert 821.10 Open fracture of unspecified part of femur 821.11 Open fracture of shaft of femur convert 821.20 Closed fracture of lower end of femur, unspecified part 821.21 Closed fracture of condyle, femoral 821.23 Closed supracondylar fracture of femur 821.29 Other closed fracture of lower end of femur 821.3 Open fracture of lower end of femur 821.30 Open fracture of lower end of femur, unspecified part 821.31 Open fracture of condyle, femoral 821.32 Open fracture of epiphysis. Lower (separation) of femur 821.33 Open supracondylar fracture of femur 821.39 Other open fracture of lower end of femur HIP AND FEMUR FRACTURES ICD10 Diagnosis codes (incident fracture - excluding subsequent encounter and sequela, and rare fractures in young children) S72.0 Fracture of head and neck of femur (all) S72.00 Fracture of unspecified part of neck of femur S72.001 Fracture of unspecified part of neck of right femur S72.001A ..... initial encounter for closed fracture S72.001B ..... initial encounter for open fracture type I or II S72.001C ..... initial encounter for open fracture type IIIA, IIIB, or IIIC S72.002 Fracture of unspecified part of neck of left femur S72.002A ..... initial encounter for closed fracture S72.002B ..... initial encounter for open fracture type I or II \$72.002C ..... initial encounter for open fracture type IIIA, IIIB, or IIIC S72.009 Fracture of unspecified part of neck of unspecified femur S72.009A ..... initial encounter for closed fracture

| S72.009B initial encounter for open fracture type I or II |
|---|
| S72.009C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.01 Unspecified intracapsular fracture of femur |
| S72.011 Unspecified intracapsular fracture of right femur |
| S72.011A initial encounter for closed fracture |
| S72.011B initial encounter for open fracture type I or II |
| S72.011C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.012 Unspecified intracapsular fracture of left femur |
| S72.012A initial encounter for closed fracture |
| S72.012B initial encounter for open fracture type I or II |
| S72.012C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.019 Unspecified intracapsular fracture of unspecified femur |
| S72.019A initial encounter for closed fracture |
| S72.019B initial encounter for open fracture type I or II |
| S72.019C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.021 Displaced fracture of epiphysis (separation) (upper) of right femur |
| S72.021A initial encounter for closed fracture |
| S72.021B initial encounter for open fracture type I or II |
| S72.021C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.022 Displaced fracture of epiphysis (separation) (upper) of left femur |
| S72.022A initial encounter for closed fracture |
| S72.022B initial encounter for open fracture type I or II |
| S72.022C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.023 Displaced fracture of epiphysis (separation) (upper) of unspecified femur |
| S72.023A initial encounter for closed fracture |
| S72.023B initial encounter for open fracture type I or II |
| S72.023C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.03 Midcervical fracture of femur |
| S72.031 Displaced midcervical fracture of right femur |
| S72.031A initial encounter for closed fracture |
| S72.031B initial encounter for open fracture type I or II |
| S72.031C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.032 Displaced midcervical fracture of left femur |
| S72.032A initial encounter for closed fracture |
| S72.032B initial encounter for open fracture type I or II |
| S72.032C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.033 Displaced midcervical fracture of unspecified femur |
| S72.033A initial encounter for closed fracture |
| S72.033B initial encounter for open fracture type I or II |
| S72.033C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.034 Nondisplaced midcervical fracture of right femur |
| S72.034A initial encounter for closed fracture |
| S72.034B initial encounter for open fracture type I or II |
| S72.034C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.035 Nondisplaced midcervical fracture of left femur |
| S72.035A initial encounter for closed fracture |
| S72.035B initial encounter for open fracture type I or II |
| S72.035C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.036 Nondisplaced midcervical fracture of unspecified femur |
| S72.036A initial encounter for closed fracture |
| S72.036B initial encounter for open fracture type I or II |
| S72.036C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.04 Fracture of base of neck of femur |
| S72.041 Displaced fracture of base of neck of right femur |
| S72.041A initial encounter for closed fracture |
| S72.041B initial encounter for open fracture type I or II |
| S72.041C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.042 Displaced fracture of base of neck of left femur |

| S72.042A initial encounter for closed fracture |
|---|
| S72.042B initial encounter for open fracture type I or II |
| S72.042C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.043 Displaced fracture of base of neck of unspecified femur |
| S72.043A initial encounter for closed fracture |
| S72.043B initial encounter for open fracture type I or II |
| S72.043C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.044 Nondisplaced fracture of base of neck of right femur |
| S72.044A initial encounter for closed fracture |
| S72.044B initial encounter for open fracture type I or II |
| S72.044C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.045 Nondisplaced fracture of base of neck of left femur |
| S72.045A initial encounter for closed fracture |
| S72.045B initial encounter for open fracture type I or II |
| S72.045C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.046 Nondisplaced fracture of base of neck of unspecified femur |
| S72.046A initial encounter for closed fracture |
| S72.046B initial encounter for open fracture type I or II |
| S72.046C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.05 Unspecified fracture of head of femur |
| S72.051 Unspecified fracture of head of right femur |
| S72.051A initial encounter for closed fracture |
| S72.051B initial encounter for open fracture type I or II |
| S72.051C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.052 Unspecified fracture of head of left femur |
| S72.052A initial encounter for closed fracture |
| S72.052B initial encounter for open fracture type I or II |
| S72.052C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.059 Unspecified fracture of head of unspecified femur |
| S72.059A initial encounter for closed fracture |
| S72.059B initial encounter for open fracture type I or II |
| S72.059C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.06 Articular fracture of head of femur |
| S72.061 Displaced articular fracture of head of right femur |
| S72.061A initial encounter for closed fracture |
| S72.061B initial encounter for open fracture type I or II |
| S72.061C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.062 Displaced articular fracture of head of left femur |
| S72.062A initial encounter for closed fracture |
| S72.062B initial encounter for open fracture type I or II |
| S72.062C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.063 Displaced articular fracture of head of unspecified femur |
| S72.063A initial encounter for closed fracture |
| S72.063B initial encounter for open fracture type I or II |
| S72.063C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.064 Nondisplaced articular fracture of head of right femur |
| S72.064A initial encounter for closed fracture |
| S72.064B initial encounter for crosed fracture type I or II |
| S72.064C initial encounter for open fracture type I IIA, IIIB, or IIIC |
| S72.065 Nondisplaced articular fracture of head of left femur S72.065A initial encounter for closed fracture |
| S72.065B initial encounter for open fracture type I or II |
| S72.065 C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.066 Nondisplaced articular fracture of head of unspecified femur |
| S72.066A initial encounter for closed fracture |
| S72.066B initial encounter for open fracture type I or II |
| S72.066C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.09 Other fracture of head and neck of femur |

| S72.091 Other fracture of head and neck of right femur |
|---|
| 572.0914 initial encounter for closed fracture |
| S72.091B initial encounter for open fracture type I or II |
| \$72.091C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.092 Other fracture of head and neck of left femur |
| \$72.092A initial encounter for closed fracture |
| S72.092B initial encounter for open fracture type I or II |
| \$72.092C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S72.099 Other fracture of head and neck of unspecified femur |
| S72.099A initial encounter for closed fracture |
| 572.0998 initial encounter for open fracture type I or II |
| 572.099C initial encounter for open fracture type IIIA, IIIB, or IIIC |
| S79.001A initial encounter for closed fracture |
| S79.002A initial encounter for closed fracture |
| S79.009A initial encounter for closed fracture |
| S79.091A initial encounter for closed fracture |
| S79.092A initial encounter for closed fracture |
| S79.099A initial encounter for closed fracture |
| S79.101A initial encounter for closed fracture |
| S79.102A initial encounter for closed fracture |
| S79.109A initial encounter for closed fracture |
| S79.191A initial encounter for closed fracture |
| S79.192A initial encounter for closed fracture |
| S79.199A initial encounter for closed fracture |
| Pathologic fracture |
| ICD9 Diagnosis Codes |
| 733.14Pathologic fracture of neck of femur |
| 733.15Pathologic fracture of other specified part of femur |
| ICDIA Discovering Codes |
| ICD10 Diagnosis Codes |
| M80 Osteoporosis with current pathological fracture |
| M80 Osteoporosis with current pathological fracture |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052A initial encounter for fracture |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, unspecified femur |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052A initial encounter for fracture M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059A initial encounter for fracture |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052A initial encounter for fracture M80.052A initial encounter for fracture M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059A initial encounter for fracture M80.059A initial encounter for fracture |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052A initial encounter for fracture M80.052A initial encounter for fracture M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059A initial encounter for fracture M80.059A initial encounter for fracture M80.059A initial encounter for fracture M80.059A initial encounter for fracture |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, right femur M80.85 Other osteoporosis with current pathological fracture, right femur M80.8510 Line osteoporosis with current pathological fracture, right femur M80.8514 initial encounter for fracture |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052A initial encounter for fracture M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059A initial encounter for fracture M80.85 Other osteoporosis with current pathological fracture, right femur M80.851 Other osteoporosis with current pathological fracture, right femur M80.852 Other osteoporosis with current pathological fracture, left femur |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.85 Other osteoporosis with current pathological fracture, right femur M80.851 A initial encounter for fracture M80.852 Other osteoporosis with current pathological fracture, left femur M80.852 Other osteoporosis with current pathological fracture, left femur M80.852 A initial encounter for fracture |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.85 Other osteoporosis with current pathological fracture, right femur M80.851 Other osteoporosis with current pathological fracture, left femur M80.852 Other osteoporosis with current pathological fracture, left femur M80.852 Other osteoporosis with current pathological fracture, left femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.850 Other osteoporosis with current pathological fracture, right femur M80.851 Age-related osteoporosis with current pathological fracture, right femur M80.851 Age-related osteoporosis with current pathological fracture, right femur M80.852 Other osteoporosis with current pathological fracture, left femur M80.852 Age-related osteoporosis with current pathological fracture, unspecified femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur |
| M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 initial encounter for fracture M80.85 Other osteoporosis with current pathological fracture, right femur M80.851 Other osteoporosis with current pathological fracture, right femur M80.851 Other osteoporosis with current pathological fracture, left femur M80.852 Other osteoporosis with current pathological fracture, left femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur |
| M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.0590 A initial encounter for fracture M80.851 Other osteoporosis with current pathological fracture, right femur M80.851 A initial encounter for fracture M80.852 Other osteoporosis with current pathological fracture, left femur M80.852 Other osteoporosis with current pathological fracture, left femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur |
| M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.0514 initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.059 Age-related osteoporosis with current pathological fracture, right femur M80.850 Other osteoporosis with current pathological fracture, right femur M80.851 Other osteoporosis with current pathological fracture, left femur M80.852 Other osteoporosis with current pathological fracture, left femur M80.852 Other osteoporosis with current pathological fracture, unspecified femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur M80.859 A initial encounter for fracture M84.4 Pathological fracture, femur and pelvis M84.451 Pathological fracture, right femur |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.0514 initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.85 Other osteoporosis with current pathological fracture, right femur M80.851 Other osteoporosis with current pathological fracture, left femur M80.852 Other osteoporosis with current pathological fracture, left femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.850 Other osteoporosis with current pathological fracture, right femur M80.851 Other osteoporosis with current pathological fracture, right femur M80.8510 Other osteoporosis with current pathological fracture, left femur M80.852 Other osteoporosis with current pathological fracture, left femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur M80.851 Other osteoporosis with current pathological fracture, initial encounter for fracture M80.451 Pathological fracture, right femur M80.451 Pathological fracture, right femur M80.452 Pathological fracture, left femur |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.85 Other osteoporosis with current pathological fracture, right femur M80.85 Other osteoporosis with current pathological fracture, right femur M80.851 A initial encounter for fracture M80.852 Other osteoporosis with current pathological fracture, left femur M80.852 A initial encounter for fracture M80.859 Other osteoporosis with current pathological fracture, unspecified femur M80.451 A initial encounter for fracture M84.451 Pathological fracture, femur and pelvis M84.451 Pathological fracture, inference and pelvis M84.451 Pathological fracture, femur and pelvis M84.452 Pathological fracture, left femur M84.452 A initial encounter for fracture |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, right femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.859 Other osteoporosis with current pathological fracture, right femur M80.851 Other osteoporosis with current pathological fracture, right femur M80.8510 Chier osteoporosis with current pathological fracture, left femur M80.852A initial encounter for fracture M80.859 Other osteoporosis with current pathological fracture, unspecified femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur M84.45 Pathological fracture, right femur M84.45 Pathological fracture, right femur M84.451 Pathological fracture, femur and pelvis M84.452 Pathological fracture, right femur M84.452 Pathological fracture, right femur M84.452 Pathological fracture, unspecified femur |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, right femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059A initial encounter for fracture M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.059 Age-related osteoporosis with current pathological fracture, right femur M80.851A initial encounter for fracture M80.851A initial encounter for fracture M80.852 Other osteoporosis with current pathological fracture, left femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur M80.859A initial encounter for fracture M80.859A initial encounter for fracture M84.45 Pathological fracture, not elsewhere classified M84.45 Pathological fracture, efmur and pelvis M84.45 Pathological fracture, efmur and pelvis M84.45 Pathological fracture, left femur M84.452 Pathological fracture, left femur M84.452 Pathological fracture, unspecified femur M84.452 Pathological fracture, unspecified femur M84.453A initial encounter for fracture M84.453A initial encounter for fracture |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.059 Age-related osteoporosis with current pathological fracture, right femur M80.059 Age-related osteoporosis with current pathological fracture, right femur M80.851 Other osteoporosis with current pathological fracture, right femur M80.851 Age-related setoporosis with current pathological fracture, left femur M80.852 Age-related osteoporosis with current pathological fracture, left femur M80.852 Age-related osteoporosis with current pathological fracture, left femur M80.859 Other osteoporosis with current pathological fracture, unspecified femur M80.859 Age-related osteoporosis with current pathological fracture, left femur M80.851 Age-related osteoporosis with current pathological fracture, femur and pelvis M84.451 Age-relotogical fracture, right femur M84.452 Pathological fracture, left femur M84.453 Pathological fracture, left femur M84.453 Pathological fracture, left femur M84.453 Pathological fracture, left femur M84.453 Pathological fracture, left, inspecified femur M84.459 Pathological fracture, left, inspecified |
| M80 Osteoporosis with current pathological fracture, femur M80.05 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.050 Age-related osteoporosis with current pathological fracture, left femur M80.051 Other osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.053 Age-related osteoporosis with current pathological fracture, left femur M80.0550 Age-related osteoporosis with current pathological fracture, unspecified femur M80.050 Age-related osteoporosis with current pathological fracture, unspecified femur M80.050 Age-related osteoporosis with current pathological fracture, unspecified femur M80.050 Age-related osteoporosis with current pathological fracture, unspecified femur M80.050 Age-related osteoporosis with current pathological fracture, remurant pathological frac |
| M80 Osteoporosis with current pathological fracture M80.05 Age-related osteoporosis with current pathological fracture, femur M80.051 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.053 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.050 Chrer osteoporosis with current pathological fracture, right femur M80.051 Chrer osteoporosis with current pathological fracture, right femur M80.052 Other osteoporosis with current pathological fracture, left femur M80.053 Age-related osteoporosis with current pathological fracture, left femur M80.0550 Age-related osteoporosis with current pathological fracture, left femur M80.0550 Age-related osteoporosis with current pathological fracture, unspecified femur M80.050 Age-related osteoporosis with current pathological fracture, unspecified femur M80.050 Age-related osteoporosis with current pathological fracture, left femur M80.050 Age-related osteoporo |
| M80 Osteoporosis with current pathological fracture, femur M80.05 Age-related osteoporosis with current pathological fracture, right femur M80.051A initial encounter for fracture M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, unspecified femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.059 Age-related osteoporosis with current pathological fracture, femur M80.050 Age-related osteoporosis with current pathological fracture, left femur M80.051 Other osteoporosis with current pathological fracture, left femur M80.052 Age-related osteoporosis with current pathological fracture, left femur M80.053 Age-related osteoporosis with current pathological fracture, left femur M80.0550 Age-related osteoporosis with current pathological fracture, unspecified femur M80.050 Age-related osteoporosis with current pathological fracture, unspecified femur M80.050 Age-related osteoporosis with current pathological fracture, unspecified femur M80.050 Age-related osteoporosis with current pathological fracture, unspecified femur M80.050 Age-related osteoporosis with current pathological fracture, remurant pathological frac |

M84.652 Pathological fracture in other disease, left femur M84.652A..... initial encounter for fracture M84.653 Pathological fracture in other disease, unspecified femur M84.653A..... initial encounter for fracture M84.659 Pathological fracture in other disease, hip, unspecified M84.659A..... initial encounter for fracture M84.7 Nontraumatic fracture, not elsewhere classified M84.75 Atypical femoral fracture M84.750A..... initial encounter for fracture M84.751 Incomplete atypical femoral fracture, right leg M84.751A..... initial encounter for fracture M84.752 Incomplete atypical femoral fracture, left leg M84.752A..... initial encounter for fracture M84.753 Incomplete atypical femoral fracture, unspecified leg M84.753A..... initial encounter for fracture M84.754 Complete transverse atypical femoral fracture, right leg M84.754A..... initial encounter for fracture M84.755 Complete transverse atypical femoral fracture, left leg M84.755A..... initial encounter for fracture M84.756 Complete transverse atypical femoral fracture, unspecified leg M84.756A..... initial encounter for fracture M84.757 Complete oblique atypical femoral fracture, right leg M84.757A..... initial encounter for fracture M84.758 Complete oblique atypical femoral fracture, left leg M84.758A..... initial encounter for fracture M84.759 Complete oblique atypical femoral fracture, unspecified leg M84.759A..... initial encounter for fracture Fracture Aftercare ICD9 Diagnosis Codes V54.13Aftercare for healing traumatic fracture of hip V54.15 Aftercare for healing traumatic fracture of upper leg Fracture Aftercare ICD10 Diagnosis Codes S72.001D Fx unsp part of nk of r femr, subs for clos fx w routn heal S72.002D Fx unsp part of nk of I femr, subs for clos fx w routn heal S72.009D Fx unsp prt of nk of unsp femr. 7thD S72.011D Unsp intracap fx right femur, subs for clos fx w routn heal S72.012D Unsp intracap fx left femur, subs for clos fx w routn heal S72.019D Unsp intracap fx unsp femur, subs for clos fx w routn heal S72.019E Unsp intracap fx unsp femr, 7thE S72.021D Disp fx of epiphy (separation) (upper) of r femr, 7thD S72.022D Disp fx of epiphy (separation) (upper) of I femr, 7thD S72.023D Disp fx of epiphy (separation) (upper) of unsp femr, 7thD S72.023E Disp fx of epiphy (separation) (upper) of unsp femr, 7thE S72.024D Nondisp fx of epiphy (separation) (upper) of r femr, 7thD S72.025D Nondisp fx of epiphy (separation) (upper) of I femr, 7thD S72.026D Nondisp fx of epiphy (separation) (upper) of unsp femr, 7thD S72.026E Nondisp fx of epiphy (separation) (upper) of unsp femr, 7thE S72.031D Displ midcervical fx r femur, subs for clos fx w routn heal S72.032D Displ midcervical fx I femur, subs for clos fx w routn heal S72.033D Displ midcervical fx unsp femr, 7thD S72.033E Displ midcervical fx unsp femr, 7thE S72.034D Nondisp midcervical fx r femr, subs for clos fx w routn heal S72.035D Nondisp midcervical fx I femr, subs for clos fx w routn heal S72.036D Nondisp midcervical fx unsp femr, 7thD S72.036E Nondisp midcervical fx unsp femr, 7thE S72.041D Disp fx of base of nk of r femr, 7thD

| S72.042D Disp fx of base of nk of I femr, 7thD | |
|---|---|
| S72.043D Disp fx of base of nk of unsp femr, 7thD | |
| S72.043E Disp fx of base of nk of unsp femr, 7thE | |
| S72.044D Nondisp fx of base of nk of r femr, 7thD | |
| S72.045D Nondisp fx of base of nk of I femr, 7thD | |
| S72.046D Nondisp fx of base of nk of unsp femr, 7thD | |
| S72.046E Nondisp fx of base of nk of unsp femr, 7thE | |
| S72.051D Unsp fx head of right femur, subs for clos fx w routn heal | |
| S72.052D Unsp fx head of left femur, subs for clos fx w routn heal | |
| S72.059D Unsp fx head of unsp femur, subs for clos fx w routn heal | |
| S72.061D Displartic fx head of r femr, subs for clos fx w routn heal | |
| S72.062D Displartic fx head of I femr, subs for clos fx w routn heal | |
| S72.063D Displ artic fx head of unsp femr, 7thD | |
| S72.064D Nondisp artic fx head of r femr, 7thD | |
| S72.065D Nondisp artic fx head of I femr, 7thD | |
| S72.066D Nondisp artic fx head of unsp femr, 7thD | |
| S72.091D Oth fx head/neck of r femur, subs for clos fx w routn heal | |
| S72.092D Oth fx head/neck of I femur, subs for clos fx w routn heal | |
| S72.099D Oth fx head/neck of unsp femr, subs for clos fx w routn heal | |
| S72.099E Oth fx head/neck of unsp femr, 7thE | |
| S72.101D Unsp trochan fx right femur, subs for clos fx w routn heal | |
| S72.102D Unsp trochan fx left femur, subs for clos fx w routn heal | |
| S72.109D Unsp trochan fx unsp femur, subs for clos fx w routn heal | |
| S72.109E Unsp trochan fx unsp femr, 7thE | |
| S72.111D Disp fx of greater trochanter of r femr, 7thD | |
| S72.112D Disp fx of greater trochanter of I femr, 7thD | |
| S72.113D Disp fx of greater trochanter of unsp femr, 7thD | |
| S72.114D Nondisp fx of greater trochanter of r femr, 7thD | |
| S72.115D Nondisp fx of greater trochanter of I femr, 7thD | |
| S72.116D Nondisp fx of greater trochanter of unsp femr, 7thD | |
| S72.121D Disp fx of less trochanter of r femr, 7thD | |
| S72.122D Disp fx of less trochanter of I femr, 7thD | |
| S72.123D Disp fx of less trochanter of unsp femr, 7thD | |
| S72.124D Nondisp fx of less trochanter of r femr, 7thD | |
| S72.125D Nondisp fx of less trochanter of I femr, 7thD | |
| S72.126D Nondisp fx of less trochanter of unsp femr, 7thD | |
| S72.131D Displayophyseal fx r femur, subs for clos fx w routh heal | |
| S72.132D Displayophyseal fx I femur, subs for clos fx w routh heal | |
| S72.133D Displ apophyseal fx unsp femr, subs for clos fx w routn heal | |
| S72.134D Nondisp apophyseal fx r femur, subs for clos fx w routh heal | |
| S72.135D Nondisp apophyseal fx I femur, subs for clos fx w routn heal S72.136D Nondisp apophyseal fx unsp femr, 7thD | |
| S72.141D Displ intertroch fx r femur, subs for clos fx w routn heal | |
| · | |
| S72.142D Displ intertroch fx I femur, subs for clos fx w routn heal S72.143D Displ intertroch fx unsp femr, subs for clos fx w routn heal | |
| S72.144D Nondisp intertroch fx r femur, subs for clos fx w routn heal | |
| S72.145D Nondisp intertroch fx l femur, subs for clos fx w routn heal<br>S72.146D Nondisp intertroch fx unsp femr, 7thD | |
| 372.1400 Nondisp intertroch ix unspreint, 7 tho | Stress fracture |
| ICD9 Diagnosis Codes | Sires ir acture |
| 733.96 Stress fracture of femoral neck | |
| 755.50 St. C55 Hactare of Terrioral fieck | |

733.97 Stress fracture of shaft of femur ICD10 diagnosis Codes (M84.3xxx Stress fracture) M84.351 Stress fracture, right femur M84.351A ..... initial encounter for fracture M84.352 Stress fracture, left femur

M84.352A ..... initial encounter for fracture

M84.353 Stress fracture, unspecified femur M84.353A ..... initial encounter for fracture M84.359 Stress fracture, hip, unspecified M84.359A ..... initial encounter for fracture HIP AND FEMUR FRACTURES ICD9 Procedure codes 78.55 Internal fixation of bone without fracture reduction, femur 79.05 Closed reduction of fracture without internal fixation, femur 79.15 Closed reduction of fracture with internal fixation, femur 79.25 Open reduction of fracture without internal fixation, femur 79.35 Open reduction of fracture with internal fixation, femur 79.65 Debridement of open fracture site, femur 815.1 Total hip replacement 815.2 Partial hip replacement HIP AND FEMUR FRACTURES ICD10 Procedure codes REPOSITION OQS6 Upper Femur, Right (ALL) OQS604Z Reposition Right Upper Femur with Internal Fixation Device, Open Approach OQS605Z Reposition Right Upper Femur with External Fixation Device, Open Approach 0QS606Z Reposition Right Upper Femur with Intramedullary Internal Fixation Device, Open Approach OQS60BZ Reposition Right Upper Femur with Monoplanar External Fixation Device, Open Approach OQS60CZ Reposition Right Upper Femur with Ring External Fixation Device, Open Approach OQS60DZ Reposition Right Upper Femur with Hybrid External Fixation Device, Open Approach 0QS60ZZ Reposition Right Upper Femur, Open Approach 0QS634Z Reposition Right Upper Femur with Internal Fixation Device, Percutaneous Approach OQS635Z Reposition Right Upper Femur with External Fixation Device, Percutaneous Approach OQS636Z Reposition Right Upper Femur with Intramedullary Internal Fixation Device, Percutaneous Approach OQS63BZ Reposition Right Upper Femur with Monoplanar External Fixation Device, Percutaneous Approach OQS63CZ Reposition Right Upper Femur with Ring External Fixation Device, Percutaneous Approach OQS63DZ Reposition Right Upper Femur with Hybrid External Fixation Device, Percutaneous Approach OQS63ZZ Reposition Right Upper Femur, Percutaneous Approach OQS644Z Reposition Right Upper Femur with Internal Fixation Device, Percutaneous Endoscopic Approach OQS645Z Reposition Right Upper Femur with External Fixation Device, Percutaneous Endoscopic Approach OQS646Z Reposition Right Upper Femur with Intramedullary Internal Fixation Device, Percutaneous Endoscopic Approach OQS64BZ Reposition Right Upper Femur with Monoplanar External Fixation Device, Percutaneous Endoscopic Approach OQS64CZ Reposition Right Upper Femur with Ring External Fixation Device, Percutaneous Endoscopic Approach OQS64DZ Reposition Right Upper Femur with Hybrid External Fixation Device, Percutaneous Endoscopic Approach OQS64ZZ Reposition Right Upper Femur, Percutaneous Endoscopic Approach OQS6XZZ Reposition Right Upper Femur, External Approach OQS7 Upper Femur, Left (ALL) OQS704Z Reposition Left Upper Femur with Internal Fixation Device, Open Approach OQS705Z Reposition Left Upper Femur with External Fixation Device, Open Approach OQS706Z Reposition Left Upper Femur with Intramedullary Internal Fixation Device, Open Approach OQS70BZ Reposition Left Upper Femur with Monoplanar External Fixation Device, Open Approach OQS70CZ Reposition Left Upper Femur with Ring External Fixation Device, Open Approach OQS70DZ Reposition Left Upper Femur with Hybrid External Fixation Device, Open Approach 0QS70ZZ Reposition Left Upper Femur, Open Approach 0QS734Z Reposition Left Upper Femur with Internal Fixation Device, Percutaneous Approach OQS735Z Reposition Left Upper Femur with External Fixation Device, Percutaneous Approach OQS736Z Reposition Left Upper Femur with Intramedullary Internal Fixation Device, Percutaneous Approach OQS73BZ Reposition Left Upper Femur with Monoplanar External Fixation Device, Percutaneous Approach OQS73CZ Reposition Left Upper Femur with Ring External Fixation Device, Percutaneous Approach OQS73DZ Reposition Left Upper Femur with Hybrid External Fixation Device, Percutaneous Approach OQS73ZZ Reposition Left Upper Femur, Percutaneous Approach OQS744Z Reposition Left Upper Femur with Internal Fixation Device, Percutaneous Endoscopic Approach 0QS745Z Reposition Left Upper Femur with External Fixation Device, Percutaneous Endoscopic Approach

0QS746Z Reposition Left Upper Femur with Intramedullary Internal Fixation Device, Percutaneous Endoscopic Approach OQS74BZ Reposition Left Upper Femur with Monoplanar External Fixation Device, Percutaneous Endoscopic Approach OQS74CZ Reposition Left Upper Femur with Ring External Fixation Device, Percutaneous Endoscopic Approach OQS74DZ Reposition Left Upper Femur with Hybrid External Fixation Device, Percutaneous Endoscopic Approach OQS74ZZ Reposition Left Upper Femur, Percutaneous Endoscopic Approach OQS7XZZ Reposition Left Upper Femur, External Approach OQS8 Femoral Shaft, Right (ALL) 0QS804Z Reposition Right Femoral Shaft with Internal Fixation Device, Open Approach 0QS805Z Reposition Right Femoral Shaft with External Fixation Device, Open Approach OQS806Z Reposition Right Femoral Shaft with Intramedullary Internal Fixation Device, Open Approach OQS80BZ Reposition Right Femoral Shaft with Monoplanar External Fixation Device, Open Approach OQS80CZ Reposition Right Femoral Shaft with Ring External Fixation Device, Open Approach OQS80DZ Reposition Right Femoral Shaft with Hybrid External Fixation Device, Open Approach OQS80ZZ Reposition Right Femoral Shaft, Open Approach OQS834Z Reposition Right Femoral Shaft with Internal Fixation Device, Percutaneous Approach OQS835Z Reposition Right Femoral Shaft with External Fixation Device, Percutaneous Approach OQS836Z Reposition Right Femoral Shaft with Intramedullary Internal Fixation Device, Percutaneous Approach OQS83BZ Reposition Right Femoral Shaft with Monoplanar External Fixation Device, Percutaneous Approach OQS83CZ Reposition Right Femoral Shaft with Ring External Fixation Device, Percutaneous Approach OQS83DZ Reposition Right Femoral Shaft with Hybrid External Fixation Device, Percutaneous Approach OQS83ZZ Reposition Right Femoral Shaft, Percutaneous Approach OQS844Z Reposition Right Femoral Shaft with Internal Fixation Device, Percutaneous Endoscopic Approach OQS845Z Reposition Right Femoral Shaft with External Fixation Device, Percutaneous Endoscopic Approach OQS846Z Reposition Right Femoral Shaft with Intramedullary Internal Fixation Device, Percutaneous Endoscopic Approach OQS84BZ Reposition Right Femoral Shaft with Monoplanar External Fixation Device, Percutaneous Endoscopic Approach OQS84CZ Reposition Right Femoral Shaft with Ring External Fixation Device, Percutaneous Endoscopic Approach OQS84DZ Reposition Right Femoral Shaft with Hybrid External Fixation Device, Percutaneous Endoscopic Approach OQS84ZZ Reposition Right Femoral Shaft, Percutaneous Endoscopic Approach OQS8XZZ Reposition Right Femoral Shaft, External Approach OQS9 Femoral Shaft, Left (ALL) OQS904Z Reposition Left Femoral Shaft with Internal Fixation Device, Open Approach OQS905Z Reposition Left Femoral Shaft with External Fixation Device, Open Approach OQS906Z Reposition Left Femoral Shaft with Intramedullary Internal Fixation Device, Open Approach OQS90BZ Reposition Left Femoral Shaft with Monoplanar External Fixation Device, Open Approach OQS90CZ Reposition Left Femoral Shaft with Ring External Fixation Device, Open Approach OQS90DZ Reposition Left Femoral Shaft with Hybrid External Fixation Device, Open Approach OQS90ZZ Reposition Left Femoral Shaft, Open Approach 0QS934Z Reposition Left Femoral Shaft with Internal Fixation Device, Percutaneous Approach 0QS935Z Reposition Left Femoral Shaft with External Fixation Device, Percutaneous Approach OQS936Z Reposition Left Femoral Shaft with Intramedullary Internal Fixation Device, Percutaneous Approach OQS93BZ Reposition Left Femoral Shaft with Monoplanar External Fixation Device, Percutaneous Approach OQS93CZ Reposition Left Femoral Shaft with Ring External Fixation Device, Percutaneous Approach OQS93DZ Reposition Left Femoral Shaft with Hybrid External Fixation Device, Percutaneous Approach OQS93ZZ Reposition Left Femoral Shaft, Percutaneous Approach OQS944Z Reposition Left Femoral Shaft with Internal Fixation Device, Percutaneous Endoscopic Approach OQS945Z Reposition Left Femoral Shaft with External Fixation Device, Percutaneous Endoscopic Approach OQS946Z Reposition Left Femoral Shaft with Intramedullary Internal Fixation Device, Percutaneous Endoscopic Approach OQS94BZ Reposition Left Femoral Shaft with Monoplanar External Fixation Device, Percutaneous Endoscopic Approach OQS94CZ Reposition Left Femoral Shaft with Ring External Fixation Device, Percutaneous Endoscopic Approach OQS94DZ Reposition Left Femoral Shaft with Hybrid External Fixation Device, Percutaneous Endoscopic Approach OQS94ZZ Reposition Left Femoral Shaft, Percutaneous Endoscopic Approach OQS9XZZ Reposition Left Femoral Shaft, External Approach OQSB4ZZ Reposition Right Lower Femur, Percutaneous Endoscopic Approach OQSBXZZ Reposition Right Lower Femur, External Approach OQSB Lower Femur, Right (ALL) OQSB04Z Reposition Right Lower Femur with Internal Fixation Device, Open Approach OQSB05Z Reposition Right Lower Femur with External Fixation Device, Open Approach OQSB06Z Reposition Right Lower Femur with Intramedullary Internal Fixation Device, Open Approach

OQSBOBZ Reposition Right Lower Femur with Monoplanar External Fixation Device, Open Approach OQSBOCZ Reposition Right Lower Femur with Ring External Fixation Device, Open Approach OQSBODZ Reposition Right Lower Femur with Hybrid External Fixation Device, Open Approach OQSBOZZ Reposition Right Lower Femur, Open Approach OQSB34Z Reposition Right Lower Femur with Internal Fixation Device, Percutaneous Approach OQSB35Z Reposition Right Lower Femur with External Fixation Device, Percutaneous Approach OQSB36Z Reposition Right Lower Femur with Intramedullary Internal Fixation Device, Percutaneous Approach OQSB3BZ Reposition Right Lower Femur with Monoplanar External Fixation Device, Percutaneous Approach OQSB3CZ Reposition Right Lower Femur with Ring External Fixation Device, Percutaneous Approach OQSB3DZ Reposition Right Lower Femur with Hybrid External Fixation Device, Percutaneous Approach OQSB3ZZ Reposition Right Lower Femur, Percutaneous Approach OQSB44Z Reposition Right Lower Femur with Internal Fixation Device, Percutaneous Endoscopic Approach OQSB45Z Reposition Right Lower Femur with External Fixation Device, Percutaneous Endoscopic Approach OQSB46Z Reposition Right Lower Femur with Intramedullary Internal Fixation Device, Percutaneous Endoscopic Approach OQSB4BZ Reposition Right Lower Femur with Monoplanar External Fixation Device, Percutaneous Endoscopic Approach OQSB4CZ Reposition Right Lower Femur with Ring External Fixation Device, Percutaneous Endoscopic Approach OQSB4DZ Reposition Right Lower Femur with Hybrid External Fixation Device, Percutaneous Endoscopic Approach OQSB4ZZ Reposition Right Lower Femur, Percutaneous Endoscopic Approach OQSBXZZ Reposition Right Lower Femur, External Approach OQSC Lower Femur, Left (all) OQSCO4Z Reposition Left Lower Femur with Internal Fixation Device, Open Approach OQSC05Z Reposition Left Lower Femur with External Fixation Device, Open Approach OQSC06Z Reposition Left Lower Femur with Intramedullary Internal Fixation Device, Open Approach OQSCOBZ Reposition Left Lower Femur with Monoplanar External Fixation Device, Open Approach OQSCOCZ Reposition Left Lower Femur with Ring External Fixation Device, Open Approach OQSCODZ Reposition Left Lower Femur with Hybrid External Fixation Device, Open Approach OQSCOZZ Reposition Left Lower Femur, Open Approach OQSC34Z Reposition Left Lower Femur with Internal Fixation Device, Percutaneous Approach OQSC35Z Reposition Left Lower Femur with External Fixation Device, Percutaneous Approach OQSC36Z Reposition Left Lower Femur with Intramedullary Internal Fixation Device, Percutaneous Approach OQSC3BZ Reposition Left Lower Femur with Monoplanar External Fixation Device, Percutaneous Approach OQSC3CZ Reposition Left Lower Femur with Ring External Fixation Device, Percutaneous Approach OQSC3DZ Reposition Left Lower Femur with Hybrid External Fixation Device, Percutaneous Approach OQSC3ZZ Reposition Left Lower Femur, Percutaneous Approach OQSC44Z Reposition Left Lower Femur with Internal Fixation Device, Percutaneous Endoscopic Approach OQSC45Z Reposition Left Lower Femur with External Fixation Device, Percutaneous Endoscopic Approach OQSC46Z Reposition Left Lower Femur with Intramedullary Internal Fixation Device, Percutaneous Endoscopic Approach OQSC4BZ Reposition Left Lower Femur with Monoplanar External Fixation Device, Percutaneous Endoscopic Approach OQSC4CZ Reposition Left Lower Femur with Ring External Fixation Device, Percutaneous Endoscopic Approach OQSC4DZ Reposition Left Lower Femur with Hybrid External Fixation Device, Percutaneous Endoscopic Approach OQSC4ZZ Reposition Left Lower Femur, Percutaneous Endoscopic Approach OQSCXZZ Reposition Left Lower Femur, External Approach INSERTION OQH6 Upper Femur, Right (ALL) 0QH604Z Insertion of Internal Fixation Device into Right Upper Femur, Open Approach OQH605Z Insertion of External Fixation Device into Right Upper Femur, Open Approach OQH606Z Insertion of Intramedullary Internal Fixation Device into Right Upper Femur, Open Approach OQH608Z Insertion of Limb Lengthening External Fixation Device into Right Upper Femur, Open Approach OQH60BZ Insertion of Monoplanar External Fixation Device into Right Upper Femur, Open Approach OQH60CZ Insertion of Ring External Fixation Device into Right Upper Femur, Open Approach OQH60DZ Insertion of Hybrid External Fixation Device into Right Upper Femur, Open Approach OQH634Z Insertion of Internal Fixation Device into Right Upper Femur, Percutaneous Approach OQH635Z Insertion of External Fixation Device into Right Upper Femur, Percutaneous Approach OQH636Z Insertion of Intramedullary Internal Fixation Device into Right Upper Femur, Percutaneous Approach OQH638Z Insertion of Limb Lengthening External Fixation Device into Right Upper Femur, Percutaneous Approach OQH63BZ Insertion of Monoplanar External Fixation Device into Right Upper Femur, Percutaneous Approach OQH63CZ Insertion of Ring External Fixation Device into Right Upper Femur, Percutaneous Approach

OQH63DZ Insertion of Hybrid External Fixation Device into Right Upper Femur, Percutaneous Approach OQH644Z Insertion of Internal Fixation Device into Right Upper Femur, Percutaneous Endoscopic Approach OQH645Z Insertion of External Fixation Device into Right Upper Femur, Percutaneous Endoscopic Approach OQH646Z Insertion of Intramedullary Internal Fixation Device into Right Upper Femur, Percutaneous Endoscopic Approach OQH648Z Insertion of Limb Lengthening External Fixation Device into Right Upper Femur, Percutaneous Endoscopic Approach OQH64BZ Insertion of Monoplanar External Fixation Device into Right Upper Femur, Percutaneous Endoscopic Approach OQH64CZ Insertion of Ring External Fixation Device into Right Upper Femur, Percutaneous Endoscopic Approach OQH64DZ Insertion of Hybrid External Fixation Device into Right Upper Femur, Percutaneous Endoscopic Approach OQHC Lower Femur, Left (all) 0QH704Z Insertion of Internal Fixation Device into Left Upper Femur, Open Approach 0QH705Z Insertion of External Fixation Device into Left Upper Femur, Open Approach OQH706Z Insertion of Intramedullary Internal Fixation Device into Left Upper Femur, Open Approach 0QH708Z Insertion of Limb Lengthening External Fixation Device into Left Upper Femur, Open Approach OQH70BZ Insertion of Monoplanar External Fixation Device into Left Upper Femur, Open Approach OQH70CZ Insertion of Ring External Fixation Device into Left Upper Femur, Open Approach OQH70DZ Insertion of Hybrid External Fixation Device into Left Upper Femur, Open Approach 0QH734Z Insertion of Internal Fixation Device into Left Upper Femur, Percutaneous Approach 0QH735Z Insertion of External Fixation Device into Left Upper Femur, Percutaneous Approach OQH736Z Insertion of Intramedullary Internal Fixation Device into Left Upper Femur, Percutaneous Approach OQH738Z Insertion of Limb Lengthening External Fixation Device into Left Upper Femur, Percutaneous Approach OQH73BZ Insertion of Monoplanar External Fixation Device into Left Upper Femur, Percutaneous Approach OQH73CZ Insertion of Ring External Fixation Device into Left Upper Femur, Percutaneous Approach OQH73DZ Insertion of Hybrid External Fixation Device into Left Upper Femur, Percutaneous Approach OQH744Z Insertion of Internal Fixation Device into Left Upper Femur, Percutaneous Endoscopic Approach OQH745Z Insertion of External Fixation Device into Left Upper Femur, Percutaneous Endoscopic Approach OQH746Z Insertion of Intramedullary Internal Fixation Device into Left Upper Femur, Percutaneous Endoscopic Approach OQH748Z Insertion of Limb Lengthening External Fixation Device into Left Upper Femur, Percutaneous Endoscopic Approach OQH74BZ Insertion of Monoplanar External Fixation Device into Left Upper Femur, Percutaneous Endoscopic Approach OQH74CZ Insertion of Ring External Fixation Device into Left Upper Femur, Percutaneous Endoscopic Approach OQH74DZ Insertion of Hybrid External Fixation Device into Left Upper Femur, Percutaneous Endoscopic Approach OQH8 Femoral Shaft, Right (all) 0QH804Z Insertion of Internal Fixation Device into Right Femoral Shaft, Open Approach 0QH805Z Insertion of External Fixation Device into Right Femoral Shaft, Open Approach OQH806Z Insertion of Intramedullary Internal Fixation Device into Right Femoral Shaft, Open Approach OQH807Z Insertion of Intramedullary Limb Lengthening Internal Fixation Device into Right Femoral Shaft, Open Approach OQH808Z Insertion of Limb Lengthening External Fixation Device into Right Femoral Shaft, Open Approach OQH80BZ Insertion of Monoplanar External Fixation Device into Right Femoral Shaft, Open Approach 0QH80CZ Insertion of Ring External Fixation Device into Right Femoral Shaft, Open Approach OQH80DZ Insertion of Hybrid External Fixation Device into Right Femoral Shaft, Open Approach 0QH834Z Insertion of Internal Fixation Device into Right Femoral Shaft, Percutaneous Approach OQH835Z Insertion of External Fixation Device into Right Femoral Shaft, Percutaneous Approach OQH836Z Insertion of Intramedullary Internal Fixation Device into Right Femoral Shaft, Percutaneous Approach OQH837Z Insertion of Intramedullary Limb Lengthening Internal Fixation Device into Right Femoral Shaft, Percutaneous Approach OQH838Z Insertion of Limb Lengthening External Fixation Device into Right Femoral Shaft, Percutaneous Approach OQH83BZ Insertion of Monoplanar External Fixation Device into Right Femoral Shaft, Percutaneous Approach OQH83CZ Insertion of Ring External Fixation Device into Right Femoral Shaft, Percutaneous Approach OQH83DZ Insertion of Hybrid External Fixation Device into Right Femoral Shaft, Percutaneous Approach OQH844Z Insertion of Internal Fixation Device into Right Femoral Shaft, Percutaneous Endoscopic Approach OQH845Z Insertion of External Fixation Device into Right Femoral Shaft, Percutaneous Endoscopic Approach OQH846Z Insertion of Intramedullary Internal Fixation Device into Right Femoral Shaft, Percutaneous Endoscopic Approach OQH847Z Insertion of Intramedullary Limb Lengthening Internal Fixation Device into Right Femoral Shaft, Percutaneous Endoscopic Approach OQH848Z Insertion of Limb Lengthening External Fixation Device into Right Femoral Shaft, Percutaneous Endoscopic Approach OQH84BZ Insertion of Monoplanar External Fixation Device into Right Femoral Shaft, Percutaneous Endoscopic Approach OQH84CZ Insertion of Ring External Fixation Device into Right Femoral Shaft, Percutaneous Endoscopic Approach OQH84DZ Insertion of Hybrid External Fixation Device into Right Femoral Shaft, Percutaneous Endoscopic Approach OQH9 Femoral Shaft, Left (all) 0QH904Z Insertion of Internal Fixation Device into Left Femoral Shaft, Open Approach OQH905Z Insertion of External Fixation Device into Left Femoral Shaft, Open Approach

0QH906Z Insertion of Intramedullary Internal Fixation Device into Left Femoral Shaft, Open Approach OQH907Z Insertion of Intramedullary Limb Lengthening Internal Fixation Device into Left Femoral Shaft, Open Approach 0QH908Z Insertion of Limb Lengthening External Fixation Device into Left Femoral Shaft, Open Approach OQH90BZ Insertion of Monoplanar External Fixation Device into Left Femoral Shaft, Open Approach 0QH90CZ Insertion of Ring External Fixation Device into Left Femoral Shaft, Open Approach OQH90DZ Insertion of Hybrid External Fixation Device into Left Femoral Shaft, Open Approach 0QH934Z Insertion of Internal Fixation Device into Left Femoral Shaft, Percutaneous Approach OQH935Z Insertion of External Fixation Device into Left Femoral Shaft, Percutaneous Approach OQH936Z Insertion of Intramedullary Internal Fixation Device into Left Femoral Shaft, Percutaneous Approach OQH937Z Insertion of Intramedullary Limb Lengthening Internal Fixation Device into Left Femoral Shaft, Percutaneous Approach OQH938Z Insertion of Limb Lengthening External Fixation Device into Left Femoral Shaft, Percutaneous Approach OQH93BZ Insertion of Monoplanar External Fixation Device into Left Femoral Shaft, Percutaneous Approach OQH93CZ Insertion of Ring External Fixation Device into Left Femoral Shaft, Percutaneous Approach OQH93DZ Insertion of Hybrid External Fixation Device into Left Femoral Shaft, Percutaneous Approach OQH944Z Insertion of Internal Fixation Device into Left Femoral Shaft, Percutaneous Endoscopic Approach OQH945Z Insertion of External Fixation Device into Left Femoral Shaft, Percutaneous Endoscopic Approach OQH946Z Insertion of Intramedullary Internal Fixation Device into Left Femoral Shaft, Percutaneous Endoscopic Approach OQH947Z Insertion of Intramedullary Limb Lengthening Internal Fixation Device into Left Femoral Shaft, Percutaneous Endoscopic Approach OQH948Z Insertion of Limb Lengthening External Fixation Device into Left Femoral Shaft, Percutaneous Endoscopic Approach OQH94BZ Insertion of Monoplanar External Fixation Device into Left Femoral Shaft, Percutaneous Endoscopic Approach OQH94CZ Insertion of Ring External Fixation Device into Left Femoral Shaft, Percutaneous Endoscopic Approach OQH94DZ Insertion of Hybrid External Fixation Device into Left Femoral Shaft, Percutaneous Endoscopic Approach OQHB Lower Femur, Right (all) OQHBO4Z Insertion of Internal Fixation Device into Right Lower Femur, Open Approach OQHB05Z Insertion of External Fixation Device into Right Lower Femur, Open Approach OQHB06Z nsertion of Intramedullary Internal Fixation Device into Right Lower Femur, Open Approach OQHBO8Z nsertion of Limb Lengthening External Fixation Device into Right Lower Femur, Open Approach OQHBOBZ Insertion of Monoplanar External Fixation Device into Right Lower Femur, Open Approach OQHBOCZ Insertion of Ring External Fixation Device into Right Lower Femur, Open Approach OQHBODZ Insertion of Hybrid External Fixation Device into Right Lower Femur, Open Approach OQHB34Z Insertion of Internal Fixation Device into Right Lower Femur, Percutaneous Approach OQHB35Z Insertion of External Fixation Device into Right Lower Femur, Percutaneous Approach OQHB36Z Insertion of Intramedullary Internal Fixation Device into Right Lower Femur, Percutaneous Approach OQHB38ZInsertion of Limb Lengthening External Fixation Device into Right Lower Femur, Percutaneous Approach OQHB3BZ Insertion of Monoplanar External Fixation Device into Right Lower Femur, Percutaneous Approach OQHB3CZ Insertion of Ring External Fixation Device into Right Lower Femur, Percutaneous Approach OQHB3DZ Insertion of Hybrid External Fixation Device into Right Lower Femur, Percutaneous Approach OQHB44Z Insertion of Internal Fixation Device into Right Lower Femur. Percutaneous Endoscopic Approach OQHB45Z Insertion of External Fixation Device into Right Lower Femur, Percutaneous Endoscopic Approach OQHB46Z Insertion of Intramedullary Internal Fixation Device into Right Lower Femur, Percutaneous Endoscopic Approach OQHB48Z Insertion of Limb Lengthening External Fixation Device into Right Lower Femur, Percutaneous Endoscopic Approach OQHB4BZ Insertion of Monoplanar External Fixation Device into Right Lower Femur, Percutaneous Endoscopic Approach OQHB4CZ Insertion of Ring External Fixation Device into Right Lower Femur, Percutaneous Endoscopic Approach OQHB4DZ Insertion of Hybrid External Fixation Device into Right Lower Femur, Percutaneous Endoscopic Approach OQHC Lower Femur, Left (all) OQHC04ZInsertion of Internal Fixation Device into Left Lower Femur, Open Approach OQHC05ZInsertion of External Fixation Device into Left Lower Femur, Open Approach OQHC06ZInsertion of Intramedullary Internal Fixation Device into Left Lower Femur, Open Approach OQHC08ZInsertion of Limb Lengthening External Fixation Device into Left Lower Femur, Open Approach OQHCOBZInsertion of Monoplanar External Fixation Device into Left Lower Femur. Open Approach OQHCOCZInsertion of Ring External Fixation Device into Left Lower Femur, Open Approach OQHCODZInsertion of Hybrid External Fixation Device into Left Lower Femur, Open Approach OQHC34ZInsertion of Internal Fixation Device into Left Lower Femur, Percutaneous Approach OQHC35ZInsertion of External Fixation Device into Left Lower Femur, Percutaneous Approach OQHC36ZInsertion of Intramedullary Internal Fixation Device into Left Lower Femur, Percutaneous Approach OQHC38ZInsertion of Limb Lengthening External Fixation Device into Left Lower Femur, Percutaneous Approach OQHC3BZInsertion of Monoplanar External Fixation Device into Left Lower Femur, Percutaneous Approach OQHC3CZInsertion of Ring External Fixation Device into Left Lower Femur, Percutaneous Approach

OQHC3DZInsertion of Hybrid External Fixation Device into Left Lower Femur, Percutaneous Approach OQHC44ZInsertion of Internal Fixation Device into Left Lower Femur, Percutaneous Endoscopic Approach OQHC45ZInsertion of External Fixation Device into Left Lower Femur, Percutaneous Endoscopic Approach  ${\tt OQHC46ZInsertion\ of\ Intramedullary\ Internal\ Fixation\ Device\ into\ Left\ Lower\ Femur,\ Percutaneous\ Endoscopic\ A}$ OQHC48ZInsertion of Limb Lengthening External Fixation Device into Left Lower Femur, Percutaneous Endoscopic OQHC4BZInsertion of Monoplanar External Fixation Device into Left Lower Femur, Percutaneous Endoscopic Appro OQHC4CZInsertion of Ring External Fixation Device into Left Lower Femur, Percutaneous Endoscopic Approach OQHC4DZInsertion of Hybrid External Fixation Device into Left Lower Femur, Percutaneous Endoscopic Approach HIP AND FEMUR FRACTURES HCPCS/CPT codes 27125Hemiarthroplasty, hip, partial (eg, femoral stem prosthesis, bipolar arthroplasty) 27130Arthroplasty, acetabular and proximal femoral prosthetic replacement (total hip arthroplasty), with or without autograft por allograft 27220Closed treatment of acetabulum (hip socket) fracture(s) 27222Closed treatment of acetabulum (hip socket) fracture(s) 27226Fracture and/or Dislocation Procedures on the Pelvis and Hip Joint 27227Fracture and/or Dislocation Procedures on the Pelvis and Hip Joint 27228Fracture and/or Dislocation Procedures on the Pelvis and Hip Joint 27230Closed treatment of femoral fracture, proximal end, neck; without manipulation 27232Closed treatment of femoral fracture, proximal end, neck; with manipulation, with or without skeletal traction 27235Percutaneous skeletal fixation of femoral fracture, proximal end, neck 27236Open treatment of femoral fracture, proximal end, neck, internal fixation or prosthetic replacement 27238Closed treatment of intertrochanteric, peritrochanteric, or subtrochanteric femoral fracture; without manipulation 27240Closed treatment of intertrochanteric, peritrochanteric, or subtrochanteric femoral fracture; with manipulation, with or without skin or skeletal traction 27245Treatment of intertrochanteric, peritrochanteric, or subtrochanteric femoral fracture 27244Treatment of intertrochanteric, peritrochanteric, or subtrochanteric femoral fracture; with plate/screw type implant, with or without cerclage 27246Closed treatment of greater trochanteric fracture, without manipulation 27248Open treatment of greater trochanteric fracture, includes internal fixation, when performed 27254Fracture Procedures on the Pelvis and Hip Joint 27267Closed treatment of femoral fracture, proximal end, head; without manipulation 27268Closed treatment of femoral fracture, proximal end, head; with manipulation 27269Open treatment of femoral fracture, proximal end, head, includes internal fixation, when performed 27500Fracture Procedures on the Femur (Thigh Region) and Knee Joint 27501Fracture Procedures on the Femur (Thigh Region) and Knee Joint

27502Fracture Procedures on the Femur (Thigh Region) and Knee Joint

27503Fracture Procedures on the Femur (Thigh Region) and Knee Joint

27506Fracture Procedures on the Femur (Thigh Region) and Knee Joint

27507Fracture Procedures on the Femur (Thigh Region) and Knee Joint

27508Fracture Procedures on the Femur (Thigh Region) and Knee Joint

27509Fracture Procedures on the Femur (Thigh Region) and Knee Joint

27510Fracture Procedures on the Femur (Thigh Region) and Knee Joint

27511Fracture Procedures on the Femur (Thigh Region) and Knee Joint

27513Fracture Procedures on the Femur (Thigh Region) and Knee Joint

27514Fracture Procedures on the Femur (Thigh Region) and Knee Joint

## Pregnancy **Diagnosis Codes** 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY **Procedure Codes** 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY

- 72.39 OTHER HIGH FORCEPS OPERATION
- 72.4 FORCEPS ROTATION OF FETAL HEAD
- 72.5 BREECH EXTRACTION
- 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.52 OTHER PARTIAL BREECH EXTRACTION
- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR
- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION
- 74.1 LOW CERVICAL CESAREAN SECTION

- 74.2 EXTRAPERITONEAL CESAREAN SECTION
- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS

Optum MarketScan

#### BEFORE PS MATCHING





The c-statistics for the propensity score model, pre-matching was 0.803. The postmatching c-statistic was 0.533

The c-statistics for the propensity score model, pre-matching was 0.714.

The postmatching c-statistic was 0.526.

#### AFTER PS MATCHING





| Variable Number of patients | Optu | m | | Marke | 4 | | POOLE | | |
|---|---|---|---|---|---|---|---|---|---|
| | T 1 10 | | • | | Marketscan | | | | 4 |
| Number of nationts | Raloxifene | Zoledronic Acid | St. Diff. | Raloxifene | Zoledronic Acid | St. Diff. | Raloxifene | Zoledronic Acid | St. Diff. |
| Demographic characteristics | 6,815 | 6,605 | | 6,694 | 13,997 | | 13,509 | 20,602 | |
| 8 I | | | | | | | | | |
| Age | 73.41 (5.90) | 74.02 (5.52) | -0.107 | 73.81 (7.06) | 75.61 (7.14) | -0.254 | 73.61 (6.50) | 75.15 (6.71) | -0.233 |
| mean (sd)<br>median [IQR] | 73.00 [68.00, 78.00] | 75.00 [69.00, 79.00] | -0.107 | 72.00 [68.00, 79.00] | 75.00 [70.00, 81.00] | -0.234 | 72.50 (6.50) | 75.13 (6.71) | -0.233 |
| Age categories | 73.00 [08.00, 78.00] | 73.00 [09.00, 79.00] | -0.550 | 72.00 [08.00, 79.00] | 73.00 [70.00, 81.00] | -0.423 | 72.30 (0.30) | 73.00 (0.71) | -0.578 |
| <70; n (%) | 2,138 (31.4%) | 1,714 (26.0%) | 0.010 | 2,366 (35.3%) | 3,498 (25.0%) | 0.019 | 4,504 (33.4%) | 5,212 (28.1%) | 0.115 |
| 70 - 74; n (%) | 1,773 (26.0%) | 1,575 (23.8%) | 0.004 | 1,604 (24.0%) | 3,134 (22.4%) | 0.003 | 3,377 (25.0%) | 4,709 (25.4%) | -0.009 |
| >= 75; n (%) | 2,904 (42.6%) | 3,316 (50.2%) | -0.011 | 2,724 (40.7%) | 7,365 (52.6%) | -0.017 | 5,628 (41.7%) | 10,681 (57.6%) | -0.322 |
| Region | _,, ( , | -, (,-) | ***** | _,,_,(,,,,,, | ,,,,,, | ***** | 2,020 (111170) | , (-,) | **** |
| Northeast; n (%) | 1,052 (15.4%) | 609 (9.2%) | 0.018 | 1,226 (18.3%) | 2,138 (15.3%) | 0.007 | 2,278 (16.9%) | 2,747 (14.8%) | 0.058 |
| South; n (%) | 2,873 (42.2%) | 2,838 (43.0%) | -0.001 | 2,225 (33.2%) | 4,693 (33.5%) | -0.001 | 5,098 (37.8%) | 7,531 (40.6%) | -0.057 |
| Midwest; n (%) | 776 (11.4%) | 1,623 (24.6%) | -0.031 | 2,183 (32.6%) | 5,245 (37.5%) | -0.008 | 2,959 (21.9%) | 6,868 (37.0%) | -0.336 |
| West; n (%) | 2,114 (31.0%) | 1,535 (23.2%) | 0.015 | 1,060 (15.8%) | 1,921 (13.8%) | 0.005 | 3,174 (23.5%) | 3,456 (18.6%) | 0.120 |
| Calendar Time | | | | | | | | | |
| Aug 2007 - Aug 2010; n (%) | 1,729 (25.4%) | 2,334 (35.3%) | -0.018 | 2,398 (35.8%) | 3,308 (23.6%) | 0.022 | 4,127 (30.6%) | 5,642 (30.4%) | 0.004 |
| Aug 2010 - Aug 2013; n (%) | 1,436 (21.1%) | 3,541 (53.6%) | -0.053 | 2,163 (32.3%) | 5,934 (42.4%) | -0.017 | 3,599 (26.7%) | 9,475 (51.1%) | -0.517 |
| Aug 2013 - Aug 2016; n (%) | 1,570 (23.0%) | 286 (4.3%) | 0.051 | 1,587 (23.7%) | 3,512 (25.1%) | -0.003 | 3,157 (23.4%) | 3,798 (20.5%) | 0.070 |
| Aug 2016 - Mar 2020; n (%) | 2,080 (30.5%) | 444 (6.7%) | 0.055 | 546 (8.2%) | 1,243 (8.9%) | -0.002 | 2,626 (19.4%) | 1,687 (9.1%) | 0.298 |
| Metropolitan Statistical Area | | | | | | | | | |
| Urban; n (%) | N/A | N/A | N/A | 5,124 (76.5%) | 10,520 (75.2%) | 0.001 | 5,122 (76.6%) | 9,932 (75.2%) | 0.002 |
| Rural; n (%) | N/A | N/A | N/A | 94 (1.4%) | 256 (1.8%) | -0.003 | 94 (1.4%) | 246 (1.9%) | -0.004 |
| Unknown/Missing; n (%) | N/A | N/A | N/A | 1,476 (22.0%) | 3,221 (23.0%) | -0.002 | 1,475 (22.0%) | 3,030 (22.9%) | -0.002 |
| General Health Related Measures | 525 (7.79/) | 500 (0.00() | 0.004 | 257 (2.00() | 000 (5.70() | 0.000 | 702 (5.00() | 1 200 (7 50/) | 0.060 |
| Smoking; n (%) | 525 (7.7%) | 588 (8.9%) | -0.004 | 257 (3.8%) | 800 (5.7%) | -0.009 | 782 (5.8%) | 1,388 (7.5%) | -0.068 |
| Alcohol/Drug abuse or dependence; n (%) | 21 (0.3%) | 15 (0.2%) | 0.002<br>0.020 | 5 (0.1%) | 22 (0.2%) | -0.003<br>-0.005 | 026 (0.2%) | 037 (0.2%) | 0.000<br>0.075 |
| Obesity or Overweight; n (%) | 770 (11.3%)<br>416 (6.1%) | 371 (5.6%)<br>277 (4.2%) | 0.020 | 277 (4.1%) | 723 (5.2%)<br>509 (3.6%) | -0.005 | 1,047 (7.8%)<br>583 (4.3%) | 1,094 (5.9%)<br>786 (4.2%) | 0.075 |
| Obesity; n (%) Overweight; n (%) | 416 (6.1%) | 115 (1.7%) | 0.008 | 167 (2.5%)<br>127 (1.9%) | 251 (1.8%) | 0.006 | 583 (4.3%) 541 (4.0%) | 366 (2.0%) | 0.003 |
| Cardiovascular Measures | 414 (0.178) | 113 (1.770) | 0.022 | 127 (1.976) | 231 (1.876) | 0.001 | 341 (4.076) | 300 (2.076) | 0.117 |
| Hypertension; n (%) | 4,171 (61.2%) | 4,326 (65.5%) | -0.005 | 3,474 (51.9%) | 8,219 (58.7%) | -0.009 | 7,645 (56.6%) | 12,545 (67.6%) | -0.228 |
| Hyperlipidemia; n (%) | 4,597 (67.5%) | 4,422 (66.9%) | 0.003 | 3,247 (48.5%) | 7,278 (52.0%) | -0.005 | 7,844 (58.1%) | 11,700 (63.1%) | -0.102 |
| Coronary artery disease (MI, angina, Coronary atherosclerosis and | | | | | | | | , , , | |
| other forms of chronic ischemic heart disease); n (%) | 857 (12.6%) | 1,130 (17.1%) | -0.012 | 813 (12.1%) | 2,486 (17.8%) | -0.015 | 1,670 (12.4%) | 3,616 (19.5%) | -0.195 |
| Old MI; n (%) | 98 (1.4%) | 157 (2.4%) | -0.007 | 49 (0.7%) | 190 (1.4%) | -0.007 | 147 (1.1%) | 347 (1.9%) | -0.066 |
| Acute MI; n (%) | 39 (0.6%) | 65 (1.0%) | -0.004 | 37 (0.6%) | 150 (1.1%) | -0.005 | 076 (0.6%) | 215 (1.2%) | -0.064 |
| ACS/unstable angina; n (%) | 53 (0.8%) | 90 (1.4%) | -0.006 | 78 (1.2%) | 213 (1.5%) | -0.003 | 131 (1.0%) | 303 (1.6%) | -0.053 |
| Stable angina; n (%) | 223 (3.3%) | 203 (3.1%) | 0.001 | 145 (2.2%) | 407 (2.9%) | -0.004 | 368 (2.7%) | 610 (3.3%) | -0.035 |
| Coronary atherosclerosis and other CHD; n (%) | 719 (10.6%) | 1,010 (15.3%) | -0.013 | 710 (10.6%) | 2,205 (15.8%) | -0.014 | 1,429 (10.6%) | 3,215 (17.3%) | -0.194 |
| History of CABG or PTCA; n (%) | 133 (2.0%) | 222 (3.4%) | -0.009 | 60 (0.9%) | 231 (1.7%) | -0.007 | 193 (1.4%) | 453 (2.4%) | -0.073 |
| Cerebrovascular disease (Stroke, TIA, Late effects); n (%) | 281 (4.1%) | 451 (6.8%) | -0.012 | 250 (3.7%) | 948 (6.8%) | -0.014 | 531 (3.9%) | 1,399 (7.5%) | -0.156 |
| Stroke (Ischemic or hemorrhagic); n (%) | 134 (2.0%) | 228 (3.5%) | -0.009 | 114 (1.7%) | 516 (3.7%) | -0.012 | 248 (1.8%) | 744 (4.0%) | -0.131 |
| TIA; n (%) | 130 (1.9%) | 230 (3.5%) | -0.010 | 129 (1.9%) | 455 (3.3%) | -0.009 | 259 (1.9%) | 685 (3.7%) | -0.109 |
| Late effects of cerebrovascular disease; n (%) | 91 (1.3%) | 128 (1.9%) | -0.005 | 57 (0.9%) | 227 (1.6%) | -0.006 | 148 (1.1%) | 355 (1.9%) | -0.066 |
| Heart Failure; n (%) | 224 (3.3%) | 373 (5.6%) | -0.011 | 218 (3.3%) | 680 (4.9%) | -0.008 | 442 (3.3%) | 1,053 (5.7%) | -0.116 |
| Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) | 480 (7.0%) | 563 (8.5%) | -0.005 | 348 (5.2%) | 1,077 (7.7%) | -0.010 | 828 (6.1%) | 1,640 (8.8%) | -0.103 |
| Atrial fibrillation and Other cardiac dysrhythmia; n (%) | 836 (12.3%) | 1,086 (16.4%) | -0.011 | 686 (10.2%) | 2,302 (16.4%) | -0.017 | 1,522 (11.3%) | 3,388 (18.3%) | -0.198 |
| Atrial fibrillation; n (%) | 385 (5.6%) | 582 (8.8%) | -0.012 | 294 (4.4%) | 1,261 (9.0%) | -0.018 | 679 (5.0%) | 1,843 (9.9%) | -0.187 |
| Other cardiac dysrhythmia; n (%) | 689 (10.1%) | 774 (11.7%) | -0.005 | 529 (7.9%) | 1,617 (11.6%) | -0.012 | 1,218 (9.0%) | 2,391 (12.9%) | -0.125 |
| Diabetes Related Measures | 1 249 (10 99/) | 1 245 (10 00/) | 0.002 | 1.025 (15.50() | 2 520 (18 10/) | 0.006 | 2 202 (17 (0/) | 2 704 (20 40/) | 0.071 |
| Diabetes with or w/o complications; n (%) | 1,348 (19.8%) | 1,245 (18.8%) | 0.002<br>0.003 | 1,035 (15.5%) | 2,539 (18.1%) | -0.006 | 2,383 (17.6%) | 3,784 (20.4%) | -0.071 |
| Diabetes mellitus without mention of complications; n (%) | 1,266 (18.6%) | 1,140 (17.3%) | | 944 (14.1%) | 2,305 (16.5%) | -0.006 | 2,210 (16.4%) | 3,445 (18.6%) | -0.058 |
| Diabetes with specified complications; n (%) | 361 (5.3%) | 402 (6.1%) | -0.003 | 230 (3.4%) | 723 (5.2%) | -0.009<br>-0.003 | 591 (4.4%) | 1,125 (6.1%) | -0.076<br>0.000 |
| Diabetes with unspecified complications; n (%) | 83 (1.2%) | 66 (1.0%) | 0.002<br>-0.002 | 36 (0.5%) | 101 (0.7%) | -0.003<br>-0.003 | 119 (0.9%) | 167 (0.9%) | -0.029 |
| Hypoglycemia; n (%) GI Conditions | 67 (1.0%) | 77 (1.2%) | -0.002 | 54 (0.8%) | 153 (1.1%) | -0.003 | 121 (0.9%) | 230 (1.2%) | -0.029 |
| Malabsorption disorders (Non-infective enteritis and colitis, other | | | | | | | | | |
| intestinal mal., operative-related disorders of the digestive | 617 (9.1%) | 947 (14.3%) | -0.015 | 667 (10.0%) | 1,797 (12.8%) | -0.008 | 1,284 (9.5%) | 2,744 (14.8%) | -0.163 |
| system); n (%) | 017 (7.170) | 777 (17.570) | 0.013 | 007 (10.070) | 1,/// (12.0/0) | -0.000 | 1,207 (7.570) | 2,/77 (17.0/0) | -0.103 |
| Non-infective enteritis and colitis; n (%) | 388 (5.7%) | 638 (9.7%) | -0.014 | 424 (6.3%) | 1,200 (8.6%) | -0.008 | 812 (6.0%) | 1,838 (9.9%) | -0.145 |
| Other intestinal malabsorption; n (%) | 39 (0.6%) | 62 (0.9%) | -0.003 | 39 (0.6%) | 134 (1.0%) | -0.004 | 078 (0.6%) | 196 (1.1%) | -0.054 |

| Intraoperative and postprocedural complications and disorders of digestive system; n (%) | 259 (3.8%) | 369 (5.6%) | -0.008 | 275 (4.1%) | 683 (4.9%) | -0.004 | 534 (4.0%) | 1,052 (5.7%) | -0.079 |
|---|---|---|---|---|---|---|---|---|---|
| Upper GI (Diseases of esophagus, stomach and duodenum); n (%) | 2,152 (31.6%) | 2,650 (40.1%) | -0.014 | 1,566 (23.4%) | 4,379 (31.3%) | -0.015 | 3,718 (27.5%) | 7,029 (37.9%) | -0.223 |
| GI bleeding; n (%) | 303 (4.4%) | 345 (5.2%) | -0.004 | 284 (4.2%) | 655 (4.7%) | -0.002 | 587 (4.3%) | 1,000 (5.4%) | -0.051 |
| Disorders of gallbladder, biliary tract and pancreas; n (%) | 225 (3.3%) | 217 (3.3%) | 0.000 | 153 (2.3%) | 467 (3.3%) | -0.006 | 378 (2.8%) | 684 (3.7%) | -0.051 |
| Rheumatic Conditions | 223 (3.370) | 217 (3.370) | 0.000 | 103 (2.570) | 107 (3.370) | 0.000 | 370 (2.070) | 001 (3.770) | 0.051 |
| Rheumatoid arthritis and other inflammatory polyarthropathies; n | | | | | | | | | |
| (%) | 40 (0.6%) | 44 (0.7%) | -0.001 | 18 (0.3%) | 137 (1.0%) | -0.009 | 058 (0.4%) | 181 (1.0%) | -0.072 |
| Osteoarthrosis; n (%) | 2,073 (30.4%) | 2,519 (38.1%) | -0.013 | 1,684 (25.2%) | 4,966 (35.5%) | -0.019 | 3,757 (27.8%) | 7,485 (40.3%) | -0.266 |
| Other rheumatic disorders (including gout); n (%) | 4,099 (60.1%) | 4,410 (66.8%) | -0.008 | 3,608 (53.9%) | 8,399 (60.0%) | -0.008 | 7,707 (57.1%) | 12,809 (69.0%) | -0.248 |
| Gout and other crystal arthropathies; n (%) | 151 (2.2%) | 135 (2.0%) | 0.001 | 69 (1.0%) | 222 (1.6%) | -0.005 | 220 (1.6%) | 357 (1.9%) | -0.023 |
| Other rheumatic disorders; n (%) | 4,052 (59.5%) | 4,388 (66.4%) | -0.009 | 3,579 (53.5%) | 8,336 (59.6%) | -0.008 | 7,631 (56.5%) | 12,724 (68.6%) | -0.252 |
| Neuro Conditions | | | | | | | | | |
| Parkinson's disease; n (%) | 26 (0.4%) | 11 (0.2%) | 0.004 | 18 (0.3%) | 30 (0.2%) | 0.002 | 044 (0.3%) | 041 (0.2%) | 0.020 |
| Alzheimer and other Dementia Disease ; n (%) | 366 (5.4%) | 480 (7.3%) | -0.008 | 256 (3.8%) | 911 (6.5%) | -0.012 | 622 (4.6%) | 1,391 (7.5%) | -0.122 |
| Seizure disorders (epilepsy); n (%) | 53 (0.8%) | 85 (1.3%) | -0.005 | 34 (0.5%) | 143 (1.0%) | -0.006 | 087 (0.6%) | 228 (1.2%) | -0.064 |
| Delirium/Psychosis; n (%) | 124 (1.8%) | 162 (2.5%) | -0.005 | 112 (1.7%) | 335 (2.4%) | -0.005 | 236 (1.7%) | 497 (2.7%) | -0.068 |
| Other Conditions | | | | | | | | | |
| Hypothyroidism; n (%) | 1,800 (26.4%) | 1,941 (29.4%) | -0.006 | 1,277 (19.1%) | 3,187 (22.8%) | -0.008 | 3,077 (22.8%) | 5,128 (27.6%) | -0.111 |
| Liver disease; n (%) | 356 (5.2%) | 227 (3.4%) | 0.009 | 191 (2.9%) | 481 (3.4%) | -0.003 | 547 (4.1%) | 708 (3.8%) | 0.015 |
| Chronic kidney disease stages I-III; n (%) | 705 (10.3%) | 485 (7.3%) | 0.010 | 322 (4.8%) | 591 (4.2%) | 0.003 | 1,027 (7.6%) | 1,076 (5.8%) | 0.072 |
| Chronic kidney disease stages IV-V, ESRD; n (%) | 201 (2.9%) | 124 (1.9%) | 0.006 | 102 (1.5%) | 149 (1.1%) | 0.004 | 303 (2.2%) | 273 (1.5%) | 0.052 |
| Premature menopause; n (%) | 7 (0.1%) | 16 (0.2%) | -0.003 | 7 (0.1%) | 28 (0.2%) | -0.003 | 014 (0.1%) | 044 (0.2%) | -0.026 |
| Oophorectomy; n (%) | 5 (0.1%) | 16 (0.2%) | -0.003 | 7 (0.1%) | 11 (0.1%) | 0.000 | 012 (0.1%) | 027 (0.1%) | 0.000 |
| COPD; n (%) | 691 (10.1%) | 1,006 (15.2%) | -0.014 | 619 (9.2%) | 1,926 (13.8%) | -0.014 | 1,310 (9.7%) | 2,932 (15.8%) | -0.184 |
| Asthma; n (%) | 563 (8.3%) | 639 (9.7%) | -0.005 | 516 (7.7%) | 1,319 (9.4%) | -0.006 | 1,079 (8.0%) | 1,958 (10.6%) | -0.090 |
| Obstructive sleep apnea; n (%) | 222 (3.3%) | 314 (4.8%) | -0.007<br>-0.008 | 173 (2.6%)<br>249 (3.7%) | 651 (4.7%)<br>734 (5.2%) | -0.011<br>-0.007 | 395 (2.9%) | 965 (5.2%) | -0.117<br>-0.099 |
| Syncope; n (%) Falls; n (%) | 249 (3.7%)<br>539 (7.9%) | 350 (5.3%)<br>640 (9.7%) | -0.008 | 152 (2.3%) | 607 (4.3%) | -0.007 | 498 (3.7%)<br>691 (5.1%) | 1,084 (5.8%)<br>1,247 (6.7%) | -0.099 |
| VTE; n (%) | 86 (1.3%) | 200 (3.0%) | -0.006 | 81 (1.2%) | 390 (2.8%) | -0.011 | 167 (1.2%) | 590 (3.2%) | -0.068 |
| Gait abnormality; n (%) | 558 (8.2%) | 802 (12.1%) | -0.012 | 422 (6.3%) | 1,352 (9.7%) | -0.011 | 980 (7.3%) | 2,154 (11.6%) | -0.137 |
| Osteopenia; n (%) | 2,470 (36.2%) | 2,435 (36.9%) | -0.012 | 1,890 (28.2%) | 3,578 (25.6%) | 0.005 | 4,360 (32.3%) | 6,013 (32.4%) | -0.147 |
| Hip and femur fractures; n (%) | 165 (2.4%) | 234 (3.5%) | -0.006 | 116 (1.7%) | 508 (3.6%) | -0.012 | 281 (2.1%) | 742 (4.0%) | -0.111 |
| Vertebral fractures; n (%) | 485 (7.1%) | 872 (13.2%) | -0.019 | 559 (8.4%) | 1,814 (13.0%) | -0.014 | 1,044 (7.7%) | 2,686 (14.5%) | -0.218 |
| Other Fractures ; n (%) | 270 (4.0%) | 327 (5.0%) | -0.005 | 220 (3.3%) | 710 (5.1%) | -0.009 | 490 (3.6%) | 1,037 (5.6%) | -0.096 |
| Combined comorbidity score, 450 days | ` / | ` / | | ` ′ | ` ′ | | ` ' | , , , | |
| mean (sd) | 0.68 (1.77) | 0.78 (1.84) | -0.055 | 0.34 (1.36) | 0.66 (1.59) | -0.216 | 0.51 (1.58) | 0.69 (1.67) | -0.111 |
| median [IQR] | 0.00 [-1.00, 1.00] | 0.00 [0.00, 2.00] | 0.000 | 0.00 [-1.00, 1.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 (1.58) | 0.00 (1.67) | 0.000 |
| Frailty Score: Empirical Version 365 days as Categories | | | | | | | | | |
| < 0.12908; n (%) | 4,286 (62.9%) | 2,288 (34.6%) | 0.041 | 3,514 (52.5%) | 4,520 (32.3%) | 0.031 | 7,800 (57.8%) | 6,808 (36.7%) | 0.432 |
| 0.12908 - 0.1631167; n (%) | 1,318 (19.3%) | 1,889 (28.6%) | -0.019 | 1,639 (24.5%) | 4,003 (28.6%) | -0.008 | 2,957 (21.9%) | 5,892 (31.8%) | -0.225 |
| >= 0.1631167; n (%) | 1,211 (17.8%) | 2,428 (36.8%) | -0.036 | 1,541 (23.0%) | 5,474 (39.1%) | -0.029 | 2,752 (20.4%) | 7,902 (42.6%) | -0.492 |
| Medication Use | | | | | | | | | |
| Use of Calcitonin (salmon); n (%) | 1 (0.0%) | 2 (0.0%) | 0.000 | 275 (4.1%) | 504 (3.6%) | 0.003 | 276 (2.0%) | 506 (2.7%) | -0.046 |
| Use of oral corticosteroids; n (%) | 1,595 (23.4%) | 1,441 (21.8%) | 0.003 | 1,652 (24.7%) | 4,305 (30.8%) | -0.012 | 3,247 (24.0%) | 5,746 (31.0%) | -0.157 |
| Use of antidepressants; n (%) | 1,511 (22.2%) | 1,704 (25.8%) | -0.007 | 1,618 (24.2%) | 4,513 (32.2%) | -0.015 | 3,129 (23.2%) | 6,217 (33.5%) | -0.230 |
| Use of anticonvulsants; n (%) | 682 (10.0%) | 761 (11.5%) | -0.005 | 702 (10.5%) | 2,161 (15.4%) | -0.014 | 1,384 (10.2%) | 2,922 (15.8%) | -0.167 |
| Use of beta blocker OR calcium channel blocker; n (%) Use of PPIs; n (%) | 1,947 (28.6%)<br>1,786 (26.2%) | 1,813 (27.4%)<br>1,883 (28.5%) | 0.002<br>-0.004 | 2,048 (30.6%)<br>1,983 (29.6%) | 4,931 (35.2%)<br>5,220 (37.3%) | -0.008<br>-0.013 | 3,995 (29.6%)<br>3,769 (27.9%) | 6,744 (36.4%)<br>7,103 (38.3%) | -0.145<br>-0.222 |
| Use of opioids; n (%) | 1,786 (26.2%) | 2,200 (33.3%) | -0.004 | 2,208 (33.0%) | 5,220 (37.3%)<br>6,037 (43.1%) | -0.013<br>-0.016 | 3,769 (27.9%)<br>4,135 (30.6%) | 8,237 (44.4%) | -0.222 |
| Use of antipsychotics; n (%) | 1,927 (28.5%) | 108 (1.6%) | -0.009 | 103 (1.5%) | 302 (2.2%) | -0.016 | 208 (1.5%) | 410 (2.2%) | -0.288 |
| Use of anxiolytics/hypnotics; n (%) | 526 (7.7%) | 601 (9.1%) | -0.001 | 719 (10.7%) | 1,682 (12.0%) | -0.003 | 1,245 (9.2%) | 2,283 (12.3%) | -0.032 |
| Use of dementia meds; n (%) | 219 (3.2%) | 232 (3.5%) | -0.003 | 192 (2.9%) | 680 (4.9%) | -0.010 | 411 (3.0%) | 912 (4.9%) | -0.100 |
| Use of antiparkinsonian meds; n (%) | 171 (2.5%) | 211 (3.2%) | -0.004 | 168 (2.5%) | 543 (3.9%) | -0.008 | 339 (2.5%) | 754 (4.1%) | -0.090 |
| Use of Benzodiazepine; n (%) | 886 (13.0%) | 686 (10.4%) | 0.008 | 1,280 (19.1%) | 3,137 (22.4%) | -0.007 | 2,166 (16.0%) | 3,823 (20.6%) | -0.119 |
| All antidiabetic medications; n (%) | 762 (11.2%) | 565 (8.6%) | 0.008 | 645 (9.6%) | 1,525 (10.9%) | -0.004 | 1,407 (10.4%) | 2,090 (11.3%) | -0.029 |
| ACEI/ARB; n (%) | 2,651 (38.9%) | 2,178 (33.0%) | 0.010 | 2,539 (37.9%) | 5,556 (39.7%) | -0.003 | 5,190 (38.4%) | 7,734 (41.7%) | -0.067 |
| Use of Anticoagulants; n (%) | 297 (4.4%) | 407 (6.2%) | -0.008 | 284 (4.2%) | 1,223 (8.7%) | -0.018 | 581 (4.3%) | 1,630 (8.8%) | -0.183 |
| Use of Amiodarone; n (%) | 41 (0.6%) | 39 (0.6%) | 0.000 | 48 (0.7%) | 146 (1.0%) | -0.003 | 089 (0.7%) | 185 (1.0%) | -0.033 |
| Digoxin; n (%) | 89 (1.3%) | 112 (1.7%) | -0.003 | 104 (1.6%) | 302 (2.2%) | -0.004 | 193 (1.4%) | 414 (2.2%) | -0.060 |
| Use of Diuretics; n (%) | 1,978 (29.0%) | 1,794 (27.2%) | 0.003 | 2,103 (31.4%) | 4,693 (33.5%) | -0.004 | 4,081 (30.2%) | 6,487 (35.0%) | -0.103 |
| Use of Aspirin; n (%) | 37 (0.5%) | 42 (0.6%) | -0.001 | 59 (0.9%) | 158 (1.1%) | -0.002 | 096 (0.7%) | 200 (1.1%) | -0.042 |
| NSAIDs (NOT including aspirin); n (%) | 1,374 (20.2%) | 1,156 (17.5%) | 0.006 | 1,314 (19.6%) | 2,998 (21.4%) | -0.004 | 2,688 (19.9%) | 4,154 (22.4%) | -0.061 |
| Hormone replace therapy; n (%) | 558 (8.2%) | 598 (9.1%) | -0.003 | 840 (12.5%) | 1,682 (12.0%) | 0.001 | 1,398 (10.4%) | 2,280 (12.3%) | -0.060 |
| Other Pressors; n (%) | 45 (0.7%) | 38 (0.6%) | 0.001 | 66 (1.0%) | 134 (1.0%) | 0.000 | 111 (0.8%) | 172 (0.9%) | -0.011 |

| Use of Statins; n (%) | 2,995 (43.9%) | 2,448 (37.1%) | 0.011 | 2,970 (44.4%) | 6,633 (47.4%) | -0.004 | 5,965 (44.2%) | 9,081 (48.9%) | -0.094 |
|---|---|---|---|---|---|---|---|---|---|
| Prior bisphosphonate use; n (%) | 1,625 (23.8%) | 1,597 (24.2%) | -0.001 | 2,397 (35.8%) | 5,368 (38.4%) | -0.004 | 4,022 (29.8%) | 6,965 (37.5%) | -0.164 |
| Healthcare Utilization Measures | 1,020 (2010/1) | 1,677 (= 11270) | | _,_, (====, | 2,222 (2211,2) | | 1,022 (271070) | *,, *** (* * | |
| Number of any prescribed drug | | | | | | | | | |
| mean (sd) | 19.17 (16.44) | 20.93 (19.56) | -0.097 | 19.38 (15.88) | 25.07 (18.78) | -0.327 | 19.27 (16.16) | 23.88 (19.01) | -0.261 |
| median [IQR] | 15.00 [7.00, 27.00] | 17.00 [4.50, 32.00] | -0.111 | 16.00 [8.00, 27.00] | 22.00 [12.00, 35.00] | -0.345 | 15.50 (16.16) | 20.56 (19.01) | -0.287 |
| Number of office visits | 15.00 [7.00, 27.00] | 17.00 [4.50, 52.00] | 0.111 | 10.00 [0.00, 27.00] | 22.00 [12.00, 33.00] | -0.545 | 15.50 (10.10) | 20.50 (17.01) | -0.207 |
| mean (sd) | 11.51 (8.82) | 14.63 (10.41) | -0.323 | 9.55 (7.33) | 12.46 (8.75) | -0.361 | 10.54 (8.12) | 13.09 (9.26) | -0.293 |
| median [IOR] | 10.00 [6.00, 15.00] | 12.00 [8.00, 19.00] | -0.207 | 8.00 [4.00, 13.00] | 11.00 [6.00, 16.00] | -0.372 | 9.01 (8.12) | 11.29 (9.26) | -0.262 |
| Number of ED visits | 10.00 [0.00, 15.00] | 12.00 [8.00, 17.00] | -0.207 | 8.00 [4.00, 15.00] | 11:00 [0:00, 10:00] | -0.572 | 7.01 (0.12) | 11.27 (7.20) | -0.202 |
| mean (sd) | 0.36 (0.84) | 0.53 (1.05) | -0.179 | 0.32 (0.82) | 0.47 (1.03) | -0.161 | 0.34 (0.83) | 0.49 (1.04) | -0.159 |
| median [IOR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 (0.83) | 0.00 (1.04) | 0.000 |
| Number of Hospitalizations | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 (0.03) | 0.00 (1.04) | 0.000 |
| mean (sd) | 0.15 (0.51) | 0.25 (0.71) | -0.162 | 0.71 (2.75) | 1.15 (3.69) | -0.135 | 0.43 (1.97) | 0.89 (3.14) | -0.175 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 (1.97) | 0.00 (3.14) | 0.000 |
| Recent hospitalization (-30 days to Index Rx date); n (%) | 52 (0.8%) | 40 (0.6%) | 0.000 | 70 (1.0%) | 88 (0.6%) | 0.004 | 122 (0.9%) | 128 (0.7%) | 0.000 |
| Old hospitalizations (-450 to -31 days); n (%) | 591 (8.7%) | 999 (15.1%) | -0.019 | 752 (11.2%) | 2,464 (17.6%) | -0.017 | 1,343 (9.9%) | 3,463 (18.7%) | -0.253 |
| Number of Endocrinologist visits | 391 (8.770) | 999 (13.1%) | -0.019 | /32 (11.276) | 2,464 (17.6%) | -0.01/ | 1,343 (9.9%) | 3,403 (18.7%) | -0.233 |
| mean (sd) | 0.17 (0.88) | 0.40 (1.32) | -0.205 | 1.64 (2.66) | 1.94 (3.23) | -0.101 | 0.90 (1.97) | 1.50 (2.82) | -0.247 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.40 (1.32) | 0.000 | 1.00 [0.00, 2.00] | 1.00 [0.00, 3.00] | 0.000 | 0.50 (1.97) | 0.71 (2.82) | -0.247 |
| Number of DXA test performed | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 1.00 [0.00, 2.00] | 1.00 [0.00, 3.00] | 0.000 | 0.30 (1.97) | 0.71 (2.82) | -0.080 |
| • | 0.70 (0.57) | 0.76 (0.54) | -0.108 | 0.49 (0.53) | 0.49 (0.54) | 0.000 | 0.60.(0.55) | 0.57 (0.54) | 0.055 |
| mean (sd) | , , | , , | | | , , | | 0.60 (0.55) | 0.57 (0.54) | |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.000 | 0.50 (0.55) | 0.29 (0.54) | 0.385 |
| Number of days of hospitalization | 1.22 (7.04) | 2 10 (0 04) | 0.006 | 0.71 (2.75) | 1.15 (2.60) | 0.125 | 1.02 (5.06) | 1.42 ((.10) | 0.066 |
| mean (sd) | 1.33 (7.94) | 2.10 (9.94) | -0.086 | 0.71 (2.75) | 1.15 (3.69) | -0.135 | 1.02 (5.96) | 1.42 (6.18) | -0.066 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 (5.96) | 0.00 (6.18) | 0.000 |
| Occurrence of basic or comprehensive metabolic blood | 5,101 (74.8%) | 5,289 (80.1%) | -0.006 | 2,173 (32.5%) | 6,380 (45.6%) | -0.021 | 7,274 (53.9%) | 11,669 (62.9%) | -0.183 |
| chemistry test; n (%) | , , , , , | | | | | | | | |
| Number of HbA1C test ordered | 0.65(4.40) | 0.50 (4.44) | 0.440 | 0.04 (0.60) | 0.00 (0.00) | | 0.44 (0.05) | 0.04 (0.05) | |
| mean (sd) | 0.67 (1.19) | 0.50 (1.11) | 0.148 | 0.21 (0.69) | 0.23 (0.75) | -0.028 | 0.44 (0.97) | 0.31 (0.87) | 0.141 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 (0.97) | 0.00 (0.87) | 0.000 |
| Occurrence of flexible Sigmoidoscopy or colonoscopy or CT | 799 (11.7%) | 882 (13.4%) | -0.005 | 848 (12.7%) | 1,879 (13.4%) | -0.002 | 1,647 (12.2%) | 2,761 (14.9%) | -0.079 |
| virtual colonoscopy; n (%) | | | | | | | | | |
| Occurrence of Mammograms; n (%) | 4,575 (67.1%) | 4,379 (66.3%) | 0.001 | 3,578 (53.5%) | 6,460 (46.2%) | 0.010 | 8,153 (60.4%) | 10,839 (58.4%) | 0.041 |
| Occurrence of Pap smear; n (%) | 1,595 (23.4%) | 1,369 (20.7%) | 0.006 | 1,557 (23.3%) | 2,228 (15.9%) | 0.017 | 3,152 (23.3%) | 3,597 (19.4%) | 0.095 |
| Flu vaccine; n (%) | 2,798 (41.1%) | 3,017 (45.7%) | -0.007 | 1,593 (23.8%) | 3,925 (28.0%) | -0.008 | 4,391 (32.5%) | 6,942 (37.4%) | -0.103 |
| Pneumococcal vaccine; n (%) | 1,705 (25.0%) | 827 (12.5%) | 0.029 | 739 (11.0%) | 1,691 (12.1%) | -0.003 | 2,444 (18.1%) | 2,518 (13.6%) | 0.123 |
| Copay for pharmacy cost (charges in U.S. \$) | | | | | | | | | |
| mean (sd) | 36.83 (46.06) | 31.00 (36.88) | 0.140 | 23.13 (25.84) | 20.45 (19.81) | 0.116 | 30.04 (37.43) | 23.49 (25.91) | 0.203 |
| median [IQR] | 24.21 [12.54, 43.97] | 22.42 [10.81, 38.90] | 0.043 | 17.50 [8.54, 30.00] | 16.00 [8.28, 27.26] | 0.065 | 20.89 (37.43) | 17.85 (25.91) | 0.094 |
| Business Type | | | | | | | | | |
| Commercial; n (%) | 1,324 (19.4%) | 1,589 (24.1%) | -0.010 | N/A | N/A | N/A | 1,324 (19.4%) | 1,589 (24.1%) | -0.010 |
| Medicare; n (%) | 5,491 (80.6%) | 5,016 (75.9%) | 0.005 | N/A | N/A | N/A | 5,491 (80.6%) | 5,016 (75.9%) | 0.005 |
| Insurance Plan Type | | | | | | | | | |
| Comprehensive; n (%) | N/A | N/A | N/A | 2,485 (37.1%) | 5,421 (38.7%) | -0.003 | 2,485 (37.1%) | 5,421 (38.7%) | -0.003 |
| HMO; n (%) | N/A | N/A | N/A | 698 (10.4%) | 1,737 (12.4%) | -0.006 | 698 (10.4%) | 1,737 (12.4%) | -0.006 |
| PPO; n (%) | N/A | N/A | N/A | 3,108 (46.4%) | 6,134 (43.8%) | 0.004 | 3,108 (46.4%) | 6,134 (43.8%) | 0.004 |
| Others; n (%) | N/A | N/A | N/A | 403 (6.0%) | 705 (5.0%) | 0.004 | 403 (6.0%) | 705 (5.0%) | 0.004 |

Optum (unmatched): https://bwh-dope.aetion.com/projects/details/1406/results/64560/result/2
Marketscan (unmatched): https://bwh-dope.aetion.com/projects/details/1407/results/64559/result/2

| Number of patients | |
|---|---|
| Number of partients 3,198 3,198 5,816 5,916 7,000 7,100 | |
| According Acc | St. Diff. |
| Sealed (19) 73.9 (16.5) 73.6 (15.7) 73.6 (15.7) 73.0 (16.0) | 014 |
| Jandson 10 Rs Arab (19-80), 78.89 7.90 (19-80), 78.89 7.90 (19-80), 78.90 7.30 (18-80), 79.90 7.30 7.30 (18-80), 79.90 7.30 7.30 (18-80), 79.90 7.30 7.30 (18-80), 79.90 7.30 7 | |
| Age entreprier* 70; n f h h h h h h h h h h h h h h h h h h | -0.0106 |
| - 70, 14% | 0.0000 |
| 10 - 72, n (%) | |
| 2 - 15, 16 1,485 (46.4%) | -0.0065 |
| Reginal | 0.0000 |
| Sombleast, 16% 277 (8.7%) 300 (0.4%) 0.0021 1.028 (1.17%) 0.0007 1.322 (1.47%) 3.77 (1.86%) 3.477 (1.86%) | 0.0060 |
| South, (%) | |
| Additional Content of the Content | 0.0000 |
| Leet at (%) | -0.0206 |
| Catendar Time* | 0.0136 |
| Aug 2017 - Aug 2010 n | 0.0099 |
| Lang 2010 - Aug 2013 a, 16% 1.311 (41.09%) 1.285 (60.2%) 0.0020 1.41.04.9%) 1.404 (0.25.1%) 0.0005 3.358 (37.3%) 3.352 (37.2% Aug 2015 a, 16%) 2.96 (2.9%) 2.775 (8.5%) 0.0020 3.14.04.9%) 1.404 (0.25.1%) 0.0020 3.14.06 (0.25.1%) 0.0020 | |
| January 2013-n (%) 1.311 (14.19%) 1.285 (40.2%) 0.0013 2.447 (55.2%) 2.067 (35.5%) 0.0005 3.358 (37.3%) 3.352 (37.2%) 2.428 (2016-Mar 2020); (%) 459 (13.7%) 459 (13.7%) 442 (13.8%) 0.0020 3.21 (9.9%) 477 (82.7%) 0.0007 960 (10.7%) 919 (10.2%) 477 (82.7%) 0.0007 960 (10.7%) 919 (10.2%) 1.285 (10.2%) | -0.0149 |
| June 2016 16 50 50 525 5 | 0.0021 |
| Lang 2016 - Mar 2020, n (%) 439 (13.7%) 442 (13.8%) 0.003 \$521 (0.9%) 477 (8.2%) 0.007 960 (10.7%) 919 (10.2%) | 0.0051 |
| Netropolitan Statistical Area* N/A N/A N/A A,395 (75.6%) 4.99 (75.5%) 0.0001 4.521 (75.6%) 4.515 (75.5%) | 0.0163 |
| Libran, n (%) | 5.0105 |
| LRuta n. (%) | 0.0001 |
| Landamown/Missing; n. (%) | 0.0000 |
| General Health Related Messares Smoking; n (%) | 0.0000 |
| Smoking: n (%) | 0.0000 |
| Alcoho/Drug abuse or dependence; n (%) | -0.0173 |
| Obesity, or Overweight, ng %9* 222 (7.9%) 233 (7.3%) 0.0022 267 (4.6%) 262 (4.5%) 0.0005 51.9 (5.8%) 4.95 (5.5%) Overweight, ng %9 158 (4.9%) 51.3 (4.8%) 0.0005 61.6.2.8%) 178 (3.1%) 0.0017 31.9 (3.5%) 31.3 (3.5%) 31.3 (3.5%) 0.0022 12.3 (2.1%) 100 (1.7%) 0.0029 231 (2.6%) 196 (2.2%) 100 (2.7%) 100 (1.7%) 0.0029 231 (2.6%) 196 (2.2%) 100 (1.7%) 0.0029 231 (2.6%) 196 (2.2%) 100 (1.7%) 0.0029 231 (2.6%) 196 (2.2%) 100 (1.7%) 0.0029 231 (2.6%) 196 (2.2%) 100 (1.7%) 100 (1.7%) 0.0029 231 (2.6%) 196 (2.2%) 100 (1.7%) | 0.0258 |
| Obesity: n (%) | 0.0238 |
| Overweight, n (%) Cardiovascular Measures | |
| Cardiovascular Measures 2,020 (63.2%) 2,032 (63.5%) -0.0004 3,125 (53.7%) 3,123 (53.7%) -0.0001 5,145 (57.1%) 5,155 (57.2% 1/50 (15.7%) | -0.0107 |
| Hypertension; n (%)* 2,020 (63.2%) 2,032 (63.5%) -0.0004 3,125 (53.7%) 3,123 (53.7%) -0.0000 5,145 (57.1%) 5,155 (57.2%) 1,157 (57.3%) 1,125 (53.7%) 2,218 (69.4%) -0.0016 2,903 (49.9%) 2,946 (50.7%) -0.0011 5,080 (56.4%) 5,164 (57.3%) 5,164 (57.3%) 1,264 (13.8%) | 0.0261 |
| Hypertpidemia; n (%)* | 0.002/ |
| Coronary artery diseases (MI, angina, Coronary atherosclerosis and other forms of chronic ischemic heart disease); n (%)* Old MI; n (%) Acute MI; n (%) Acut | -0.0020 |
| other forms of chronic ischemic heart disease); n (%)* 56 (1.8%) 56 (2.2%) -0.0028 49 (0.8%) 58 (1.0%) -0.0021 105 (1.2%) 127 (1.4%) Acute Mi; n (%) 22 (0.7%) 28 (0.9%) -0.0022 32 (0.6%) 37 (0.6%) 0.0000 0.54 (0.6%) 065 (0.7%) ACS (unstable angina; n (%) 37 (1.2%) 37 (1.2%) 37 (1.2%) 37 (1.2%) 37 (1.2%) 40 (1.1%) 0.0009 107 (1.2%) 097 (1.1%) 40 (1.1%) 0.0009 107 (1.2%) 097 (1.1%) 0.0009 107 (1.2%) 0.0009 1.098 (12.2%) 1.102 (1.2%) 1.102 (1.2 | -0.0182 |
| Old MI; n (%) | 0.0029 |
| Acute MI; n (%) | 0.017 |
| ACS/unstable angin; n (%) 37 (1.2%) 33 (1.0%) 0.0019 70 (1.2%) 64 (1.1%) 0.0009 107 (1.2%) 0.97 (1.1%) Stable angin; n (%) 107 (3.3%) 96 (3.0%) 0.0017 134 (2.3%) 140 (2.4%) -0.0007 241 (2.7%) 236 (2.6%) 200 (2.2%) 427 (13.4%) 416 (13.0%) 0.0011 671 (11.5%) 686 (11.8%) -0.0009 1.098 (12.2%) 1.102 | -0.0177 |
| Stable angina; n (%) | -0.0124 |
| Coronary atherosclerosis and other CHD; n (%) | 0.0094 |
| History of CABG or PTCA; n (%) 75 (2.3%) 81 (2.5%) -0.0013 57 (1.0%) 70 (1.2%) -0.0019 132 (1.5%) 151 (1.7%) Cerebrovascular disease (Stroke, TIA, Late effects); n (%)* 162 (5.1%) 170 (5.3%) -0.0009 241 (4.1%) 241 (4.1%) 0.0000 403 (4.5%) 411 (4.6%) 411 (4.6%) 170 (5.3%) -0.0019 125 (2.1%) 129 (2.2%) -0.0021 192 (2.1%) 225 (2.5%) 141 (4.6%) -0.0019 125 (2.1%) 119 (2.0%) 0.0007 197 (2.2%) 201 (2.2%) 22% 22% 22% -0.0021 192 (2.1%) 225 (2.5%) 22.5% 22 | 0.0062 |
| Cerebrovascular disease (Stroke, TIA, Late effects); n (%)* 162 (5.1%) 170 (5.3%) -0.0009 241 (4.1%) 241 (4.1%) 0.0000 403 (4.5%) 411 (4.6%) Stroke (Ischemic or hemorrhagic); n (%) 79 (2.5%) 96 (3.0%) -0.0030 113 (1.9%) 129 (2.2%) -0.0021 192 (2.1%) 225 (2.5%) 225 (2.5%) 225 (2.5%) 119 (2.0%) 0.0007 197 (2.2%) 201 (2.2%) 226 (2.5%) 228 (2.6%) -0.0019 225 (2.1%) 119 (2.0%) 0.0007 197 (2.2%) 201 | 0.0000 |
| Stroke (Ischemic or hemorrhagic); n (%) TIA; n (%) Late effects of cerebrovascular disease; n (%) Late effects of cerebrovascular disease; n (%) Lear Failure; n (%)* Peripheral Vascular Disease (PVD) or PVD Surgery; n (%)* Atrial fibrillation and Other cardiac dysrhythmia; n (%)* Atrial fibrillation; n (%) Other cardiac dysrhythmia; n (%) Diabetes with or w/o complications; n (%) Diabetes with or sw/o complications; n (%) Diabetes with unspecified complications; n (%) TIA; n (%) Possible of the first of the | -0.0159 |
| TIA; n (%) Late effects of cerebrovascular disease; n (%) Heart Failure; n (%)* Feripheral Vascular Disease (PVD) or PVD Surgery; n (%)* Atrial fibrillation and Other cardiac dysrhythmia; n (%)* Atrial fibrillation; n (%) Other cardiac dysrhythmia; n (%) Diabetes Related Measures Diabetes with or w/o complications; n (%) Diabetes with unspecified com | -0.0048 |
| Late effects of cerebrovascular disease; n (%) Heart Failure; n (%)* Peripheral Vascular Disease (PVD) or PVD Surgery; n (%)* Atrial fibrillation and Other cardiac dysrhythmia; n (%)* Atrial fibrillation; n (%) Atrial fibrillation; n (%) Atrial fibrillation in (%) Atrial fibrillation; n (%) Atrial fibrillation of the cardiac dysrhythmia; n (%)* Atrial fibrillation; n (%) Diabetes Related Measures Diabetes with or w/o complications; n (%)* Diabetes with or w/o complications; n (%)* Diabetes with or w/o complications; n (%) Diabetes with unspecified complications; n (%) Diabetes with unspecified complications; n (%) Diabetes with unspecified complications; n (%) Atrial fibrillation; n (%) Attrial fibrillatio | -0.0267 |
| Heart Failure; n (%)* Peripheral Vascular Disease (PVD) or PVD Surgery; n (%)* Atrial fibrillation and Other cardiac dysrhythmia; n (%)* Atrial fibrillation; n (%) Atrial fibrillation; n (%) Atrial fibrillation; n (%) Atrial fibrillation; n (%) Atrial fibrillation; n (%) Diabetes Related Measures Diabetes with or w/o complications; n (%) Diabetes with specified complications; n (%) Diabetes with specified complications; n (%) Diabetes with unspecified complications; n (%) Diabetes with un | 0.0000 |
| Peripheral Vascular Disease (PVD) or PVD Surgery; n (%)* Atrial fibrillation and Other cardiac dysrhythmia; n (%)* 446 (13.9%) 445 (13.9%) 0.0018 333 (5.7%) 315 (5.4%) 0.0013 576 (6.4%) 542 (6.0%) 542 (6.0%) 542 (6.0%) 543 (1.1.5%) 0.0000 657 (11.3%) 671 (11.5%) 0.0006 1,103 (12.2%) 1,116 (12.4%) 1,116 (12.4% | 0.0192 |
| Atrial fibrillation and Other cardiac dysrhythmia; n (%)* Atrial fibrillation; n (%) Other cardiac dysrhythmia; n (%)* Diabetes Related Measures Diabetes with or w/o complications; n (%) Diabetes with unspecified comp | 0.0105 |
| Atrial fibrillation; n (%) Other cardiac dysrhythmia; n (%) Diabetes Related Measures Diabetes with or w/o complications; n (%) Diabetes with unspecified complication | 0.0166 |
| Other cardiac dysrhythmia; n (%) Diabetes Related Measures Diabetes with or w/o complications; n (%)* Diabetes with specified complications; n (%) Diabetes with unspecified complications; n (%) Hypoglycemia; n (%) GI Conditions 346 (10.8%) 334 (10.4%) 344 (10.4%) 344 | -0.0061 |
| Diabetes Related Measures Complete Related Measures Diabetes with or w/o complications; n (%)* 614 (19.2%) 635 (19.9%) -0.0016 937 (16.1%) 916 (15.7%) 0.0010 1,551 (17.2%) 1,435 (15.9%) 1,435 ( | -0.0298 |
| Diabetes with or w/o complications; n (%)* Diabetes with or w/o complications; n (%)* Diabetes mellitus without mention of complications; n (%) Diabetes mellitus without mention of complications; n (%) Diabetes with specified complications; n (%) Diabetes with unspecified complications; n (%) Diabetes with unsp | 0.0069 |
| Diabetes mellitus without mention of complications; n (%) Diabetes with specified complications; n (%) Diabetes with unspecified complications; n (%) Diabetes with un | |
| Diabetes mellitus without mention of complications; n (%) Diabetes with specified complications; n (%) Diabetes with unspecified complications; n (%) Diabetes with un | 0.0000 |
| Diabetes with specified complications; n (%) $180 (5.6\%)$ $192 (6.0\%)$ $-0.0017$ $215 (3.7\%)$ $219 (3.8\%)$ $-0.0005$ $395 (4.4\%)$ $411 (4.6\%)$ Diabetes with unspecified complications; n (%) $35 (1.1\%)$ $34 (1.1\%)$ $0.0000$ $32 (0.6\%)$ $36 (0.6\%)$ $0.0000$ $067 (0.7\%)$ $070 (0.8\%)$ Hypoglycemia; n (%) $42 (1.3\%)$ $40 (1.3\%)$ $0.0000$ $52 (0.9\%)$ $44 (0.8\%)$ $0.0011$ $094 (1.0\%)$ $084 (0.9\%)$ GI Conditions | -0.0027 |
| Diabetes with unspecified complications; n (%) $35 (1.1\%)$ $34 (1.1\%)$ $0.0000$ $32 (0.6\%)$ $36 (0.6\%)$ $0.0000$ $067 (0.7\%)$ $070 (0.8\%)$ Hypoglycemia; n (%) $42 (1.3\%)$ $40 (1.3\%)$ $0.0000$ $52 (0.9\%)$ $44 (0.8\%)$ $0.0011$ $094 (1.0\%)$ $084 (0.9\%)$ GI Conditions | -0.0096 |
| Hypoglycemia; n (%) 42 (1.3%) 40 (1.3%) 0.0000 52 (0.9%) 44 (0.8%) 0.0011 094 (1.0%) 084 (0.9%) GI Conditions | -0.0116 |
| GI Conditions | 0.0103 |
| | 0.0103 |
| intestinal mal., operative-related disorders of the digestive 363 (11.4%) 361 (11.3%) 0.0003 605 (10.4%) 625 (10.7%) -0.0009 968 (10.7%) 986 (10.9%) | -0.0064 |
| system); n (%)* | -0.0064 |
| System); n (%)* Non-infective enteritis and colitis; n (%) 230 (7.2%) 237 (7.4%) -0.0007 390 (6.7%) 387 (6.7%) 0.0000 620 (6.9%) 624 (6.9%) | 0.0000 |

| ī | • | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Other intestinal malabsorption; n (%) | 16 (0.5%) | 21 (0.7%) | -0.0026 | 37 (0.6%) | 50 (0.9%) | -0.0035 | 053 (0.6%) | 071 (0.8%) | -0.0240 |
| Intraoperative and postprocedural complications and disorders of digestive system; n (%) | 159 (5.0%) | 146 (4.6%) | 0.0018 | 248 (4.3%) | 263 (4.5%) | -0.0010 | 407 (4.5%) | 409 (4.5%) | 0.0000 |
| Upper GI (Diseases of esophagus, stomach and duodenum); n | | | | | | | | | |
| (%)* | 1,141 (35.7%) | 1,138 (35.6%) | 0.0002 | 1,466 (25.2%) | 1,430 (24.6%) | 0.0012 | 2,607 (28.9%) | 2,568 (28.5%) | 0.0088 |
| GI bleeding; n (%)* | 161 (5.0%) | 160 (5.0%) | 0.0000 | 252 (4.3%) | 269 (4.6%) | -0.0014 | 413 (4.6%) | 429 (4.8%) | -0.0095 |
| Disorders of gallbladder, biliary tract and pancreas; n (%)* | 87 (2.7%) | 88 (2.8%) | -0.0006 | 145 (2.5%) | 148 (2.5%) | 0.0000 | 232 (2.6%) | 236 (2.6%) | 0.0000 |
| Rheumatic Conditions | ` / | ` / | | ` / | ` ′ | | , , | ` / | |
| Rheumatoid arthritis and other inflammatory polyarthropathies; n | 16 (0.5%) | 28 (0.9%) | -0.0048 | 18 (0.3%) | 48 (0.8%) | -0.0067 | 034 (0.4%) | 076 (0.8%) | -0.0518 |
| (%) | ` ' | ` ' | | | ` ' | | ` ´ | ` ´ | |
| Osteoarthrosis; n (%)* | 1,087 (34.0%) | 1,111 (34.7%) | -0.0012 | 1,603 (27.6%) | 1,636 (28.1%) | -0.0009 | 2,690 (29.8%) | 2,747 (30.5%) | -0.0153 |
| Other rheumatic disorders (including gout); n (%)* | 2,019 (63.1%) | 2,045 (63.9%) | -0.0010 | 3,198 (55.0%) | 3,248 (55.8%) | -0.0011 | 5,217 (57.9%) | 5,293 (58.7%) | -0.0162 |
| Gout and other crystal arthropathies; n (%) | 70 (2.2%) | 55 (1.7%) | 0.0036 | 65 (1.1%) | 62 (1.1%) | 0.0000 | 135 (1.5%) | 117 (1.3%) | 0.0170 |
| Other rheumatic disorders; n (%) Neuro Conditions | 1,999 (62.5%) | 2,033 (63.6%) | -0.0014 | 3,170 (54.5%) | 3,225 (55.5%) | -0.0014 | 5,169 (57.3%) | 5,258 (58.3%) | -0.0202 |
| Parkinson's disease; n (%) | 8 (0.3%) | 6 (0.2%) | 0.0020 | 18 (0.3%) | 10 (0.2%) | 0.0020 | 026 (0.3%) | 016 (0.2%) | 0.0200 |
| Alzheimer and other Dementia Disease ; n (%)* | 193 (6.0%) | 189 (5.9%) | 0.0020 | 253 (4.4%) | 257 (4.4%) | 0.0020 | 446 (4.9%) | 446 (4.9%) | 0.0000 |
| Seizure disorders (epilepsy); n (%) | 29 (0.9%) | 36 (1.1%) | -0.0020 | 31 (0.5%) | 41 (0.7%) | -0.0026 | 060 (0.7%) | 077 (0.9%) | -0.0225 |
| Delirium/Psychosis; n (%) | 64 (2.0%) | 59 (1.8%) | 0.0015 | 109 (1.9%) | 84 (1.4%) | 0.0039 | 173 (1.9%) | 143 (1.6%) | 0.0229 |
| Other Conditions | . (, | () | | ( , | . ( , | | (, | , | |
| Hypothyroidism; n (%)* | 900 (28.1%) | 933 (29.2%) | -0.0021 | 1,179 (20.3%) | 1,164 (20.0%) | 0.0007 | 2,079 (23.1%) | 2,097 (23.3%) | -0.0047 |
| Liver disease; n (%)* | 109 (3.4%) | 121 (3.8%) | -0.0021 | 175 (3.0%) | 164 (2.8%) | 0.0012 | 284 (3.2%) | 285 (3.2%) | 0.0000 |
| Chronic kidney disease stages I-III; n (%)* | 284 (8.9%) | 276 (8.6%) | 0.0010 | 284 (4.9%) | 272 (4.7%) | 0.0009 | 568 (6.3%) | 548 (6.1%) | 0.0083 |
| Chronic kidney disease stages IV-V, ESRD; n (%) | 103 (3.2%) | 70 (2.2%) | 0.0061 | 89 (1.5%) | 55 (0.9%) | 0.0055 | 192 (2.1%) | 125 (1.4%) | 0.0534 |
| Premature menopause; n (%) | 3 (0.1%) | 7 (0.2%) | -0.0026 | 5 (0.1%) | 10 (0.2%) | -0.0026 | 008 (0.1%) | 017 (0.2%) | -0.0258 |
| Oophorectomy; n (%) | 3 (0.1%) | 5 (0.2%) | -0.0026 | 7 (0.1%) | 3 (0.1%) | 0.0000 | 010 (0.1%) | 008 (0.1%) | 0.0000 |
| COPD; n (%)* | 411 (12.9%) | 401 (12.5%) | 0.0011 | 584 (10.0%) | 594 (10.2%) | -0.0006 | 995 (11.0%) | 995 (11.0%) | 0.0000 |
| Asthma; n (%)* | 294 (9.2%)<br>123 (3.8%) | 300 (9.4%)<br>125 (3.9%) | -0.0007<br>-0.0005 | 461 (7.9%)<br>171 (2.9%) | 490 (8.4%)<br>152 (2.6%) | -0.0018<br>0.0018 | 755 (8.4%)<br>294 (3.3%) | 790 (8.8%)<br>277 (3.1%) | -0.0143<br>0.0114 |
| Obstructive sleep apnea; n (%)*<br>Syncope; n (%)* | 131 (4.1%) | 139 (4.3%) | -0.0003 | 236 (4.1%) | 236 (4.1%) | 0.0018 | 367 (4.1%) | 375 (4.2%) | -0.0050 |
| Falls; n (%)* | 266 (8.3%) | 272 (8.5%) | -0.0010 | 146 (2.5%) | 157 (2.7%) | -0.0012 | 412 (4.6%) | 429 (4.8%) | -0.0030 |
| VTE; n (%) | 47 (1.5%) | 72 (2.3%) | -0.0058 | 78 (1.3%) | 119 (2.0%) | -0.0012 | 125 (1.4%) | 191 (2.1%) | -0.0534 |
| Gait abnormality; n (%)* | 282 (8.8%) | 305 (9.5%) | -0.0023 | 405 (7.0%) | 373 (6.4%) | 0.0023 | 687 (7.6%) | 678 (7.5%) | 0.0038 |
| Osteopenia; n (%)* | 1,200 (37.5%) | 1,203 (37.6%) | -0.0002 | 1,585 (27.3%) | 1,626 (28.0%) | -0.0013 | 2,785 (30.9%) | 2,829 (31.4%) | -0.0108 |
| Hip and femur fractures; n (%)* | 86 (2.7%) | 98 (3.1%) | -0.0023 | 113 (1.9%) | 122 (2.1%) | -0.0014 | 199 (2.2%) | 220 (2.4%) | -0.0133 |
| Vertebral fractures; n (%)* | 298 (9.3%) | 304 (9.5%) | -0.0007 | 543 (9.3%) | 527 (9.1%) | 0.0007 | 841 (9.3%) | 831 (9.2%) | 0.0035 |
| Other Fractures; n (%)* | 141 (4.4%) | 142 (4.4%) | 0.0000 | 206 (3.5%) | 206 (3.5%) | 0.0000 | 347 (3.8%) | 348 (3.9%) | -0.0052 |
| Combined comorbidity score, 450 days* | | | | | | | | | |
| mean (sd) | 0.70 (1.83) | 0.68 (1.82) | 0.0110 | 0.40 (1.40) | 0.40 (1.37) | 0.0000 | 0.51 (1.57) | 0.50 (1.54) | 0.0064 |
| median [IQR] | 0.00 [-1.00, 1.00] | 0.00 [-1.00, 1.00] | 0.0000 | 0.00 [-1.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 (1.57) | 0.00 (1.54) | 0.0000 |
| Frailty Score: Empirical Version 365 days as Categories*< 0.12908; n (%) | 1,492 (46.7%) | 1,502 (47.0%) | -0.0004 | 2,738 (47.1%) | 2,740 (47.1%) | 0.0000 | 4,230 (46.9%) | 4,242 (47.1%) | -0.0040 |
| | 866 (27.1%) | 846 (26.5%) | 0.0012 | 1,570 (27.0%) | 1,563 (26.9%) | 0.0000 | 2,436 (27.0%) | 2,409 (26.7%) | 0.0068 |
| >= 0.1631167; n (%) | 840 (26.3%) | 850 (26.6%) | -0.0006 | 1,508 (25.9%) | 1,513 (26.0%) | -0.0002 | 2,348 (26.0%) | 2,363 (26.2%) | -0.0046 |
| Medication Use | 0.10 (=0.070) | () | | -, (=,-) | -, (=, | | _,,,,, | =,= ++ (= ++= ++) | |
| Use of Calcitonin (salmon); n (%) | 1 (0.0%) | 0 (0.0%) | 0.0000 | 243 (4.2%) | 213 (3.7%) | 0.0025 | 244 (2.7%) | 213 (2.4%) | 0.0190 |
| Use of oral corticosteroids; n (%)* | 779 (24.4%) | 770 (24.1%) | 0.0006 | 1,542 (26.5%) | 1,540 (26.5%) | 0.0000 | 2,321 (25.7%) | 2,310 (25.6%) | 0.0023 |
| Use of antidepressants; n (%)* | 836 (26.1%) | 821 (25.7%) | 0.0008 | 1,522 (26.2%) | 1,542 (26.5%) | -0.0006 | 2,358 (26.2%) | 2,363 (26.2%) | 0.0000 |
| Use of anticonvulsants; n (%)* | 353 (11.0%) | 387 (12.1%) | -0.0032 | 669 (11.5%) | 689 (11.8%) | -0.0009 | 1,022 (11.3%) | 1,076 (11.9%) | -0.0187 |
| Use of beta blocker OR calcium channel blocker; n (%)* | 1,013 (31.7%) | 1,009 (31.6%) | 0.0002 | 1,855 (31.9%) | 1,884 (32.4%) | -0.0009 | 2,868 (31.8%) | 2,893 (32.1%) | -0.0064 |
| Use of PPIs; n (%)* | 968 (30.3%) | 962 (30.1%) | 0.0004 | 1,845 (31.7%) | 1,863 (32.0%) | -0.0005 | 2,813 (31.2%) | 2,825 (31.3%) | -0.0022 |
| Use of opioids; n (%)* | 1,100 (34.4%) | 1,111 (34.7%) | -0.0005 | 2,080 (35.8%) | 2,074 (35.7%) | 0.0002 | 3,180 (35.3%) | 3,185 (35.3%) | 0.0000 |
| Use of antipsychotics; n (%)* | 58 (1.8%) | 56 (1.8%) | 0.0000<br>0.0007 | 97 (1.7%) | 86 (1.5%)<br>660 (11.3%) | 0.0016<br>0.0000 | 155 (1.7%)<br>957 (10.6%) | 142 (1.6%) | 0.0079 |
| Use of anxiolytics/hypnotics; n (%)* Use of dementia meds; n (%)* | 301 (9.4%)<br>109 (3.4%) | 293 (9.2%) | -0.0016 | 656 (11.3%)<br>188 (3.2%) | 200 (3.4%) | -0.0011 | 297 (3.3%) | 953 (10.6%)<br>317 (3.5%) | 0.0000<br>-0.0110 |
| Use of antiparkinsonian meds; n (%)* | 109 (3.4%) | 117 (3.7%)<br>105 (3.3%) | -0.0016 | 188 (3.2%) | 156 (2.7%) | 0.0001 | 260 (2.9%) | 261 (2.9%) | 0.0000 |
| Use of Benzodiazepine; n (%)* | 403 (12.6%) | 402 (12.6%) | 0.0000 | 1,192 (20.5%) | 1,196 (20.6%) | -0.0002 | 1,595 (17.7%) | 1,598 (17.7%) | 0.0000 |
| All antidiabetic medications; n (%)* | 341 (10.7%) | 351 (11.0%) | -0.0009 | 589 (10.1%) | 583 (10.0%) | 0.0003 | 930 (10.3%) | 934 (10.4%) | -0.0033 |
| ACEI/ARB; n (%)* | 1,218 (38.1%) | 1,241 (38.8%) | -0.0011 | 2,250 (38.7%) | 2,256 (38.8%) | -0.0002 | 3,468 (38.5%) | 3,497 (38.8%) | -0.0062 |
| Use of Anticoagulants; n (%)* | 176 (5.5%) | 183 (5.7%) | -0.0008 | 282 (4.8%) | 315 (5.4%) | -0.0027 | 458 (5.1%) | 498 (5.5%) | -0.0179 |
| Use of Amiodarone; n (%) | 25 (0.8%) | 19 (0.6%) | 0.0024 | 48 (0.8%) | 37 (0.6%) | 0.0024 | 073 (0.8%) | 056 (0.6%) | 0.0240 |
| Digoxin; n (%) | 52 (1.6%) | 58 (1.8%) | -0.0015 | 97 (1.7%) | 92 (1.6%) | 0.0008 | 149 (1.7%) | 150 (1.7%) | 0.0000 |
| Use of Diuretics; n (%)* | 1,021 (31.9%) | 1,041 (32.6%) | -0.0012 | 1,865 (32.1%) | 1,857 (31.9%) | 0.0004 | 2,886 (32.0%) | 2,898 (32.1%) | -0.0021 |
| Use of Aspirin; n (%) | 25 (0.8%) | 21 (0.7%) | 0.0012 | 55 (0.9%) | 56 (1.0%) | -0.0010 | 080 (0.9%) | 077 (0.9%) | 0.0000 |

| 651 (20.4%)<br>315 (9.8%)<br>23 (0.7%)<br>,427 (44.6%)<br>746 (23.3%) | 643 (20.1%)<br>318 (9.9%)<br>16 (0.5%)<br>1,443 (45.1%)<br>847 (26.5%) | 0.0007<br>-0.0003<br>0.0026<br>-0.0007<br>-0.0064 | 1,198 (20.6%)<br>743 (12.8%)<br>64 (1.1%)<br>2,677 (46.0%)<br>2,079 (35.7%) | 1,155 (19.9%)<br>751 (12.9%)<br>66 (1.1%)<br>2,656 (45.7%) | 0.0016<br>-0.0003<br>0.0000<br>0.0004 | 1,849 (20.5%)<br>1,058 (11.7%)<br>087 (1.0%)<br>4,104 (45.5%) | 1,798 (19.9%)<br>1,069 (11.9%)<br>082 (0.9%)<br>4,099 (45.5%) | 0.0149<br>-0.0062<br>0.0103<br>0.0000 |
|---|---|---|---|---|---|---|---|---|
| 23 (0.7%)<br>,427 (44.6%)<br>746 (23.3%) | 16 (0.5%)<br>1,443 (45.1%) | 0.0026<br>-0.0007 | 64 (1.1%)<br>2,677 (46.0%) | 66 (1.1%)<br>2,656 (45.7%) | 0.0000 | 087 (1.0%) | 082 (0.9%) | 0.0103 |
| ,427 (44.6%)<br>746 (23.3%) | 1,443 (45.1%) | -0.0007 | 2,677 (46.0%) | 2,656 (45.7%) | | · / | · / | |
| 746 (23.3%) | | | | | 0.0004 | 4,104 (45.5%) | 4 099 (45 5%) | 0.0000 |
| | 847 (26.5%) | -0.0064 | 2,079 (35.7%) | 2.246 (20.60/) | | | | |
| 2.08 (18.32) | | | | 2,246 (38.6%) | -0.0048 | 2,825 (31.3%) | 3,093 (34.3%) | -0.0639 |
| 2.08 (18.32) | | | | | | | | |
| 2.08 (18.32) | | | | | | | | |
| | 21.98 (16.47) | 0.0057 | 20.71 (16.23) | 20.85 (15.42) | -0.0088 | 21.20 (17.00) | 21.25 (15.80) | -0.0030 |
| 00 [8.00, 31.00] | 18.00 [10.00, 30.00] | 0.0000 | 17.00 [9.00, 28.00] | 18.00 [10.00, 28.00] | -0.0632 | 17.35 (17.00) | 18.00 (15.80) | -0.0396 |
| 12.76 (9.40) | 12.86 (8.99) | -0.0109 | 10.14 (7.52) | 10.11 (7.03) | 0.0041 | 11.07 (8.24) | 11.09 (7.78) | -0.0025 |
| 00 [6.00, 17.00] | 11.00 [7.00, 16.25] | -0.1087 | 9.00 [5.00, 14.00] | 9.00 [5.00, 13.00] | 0.0000 | 9.35 (8.24) | 9.71 (7.78) | -0.0449 |
| 0.42 (0.91) | 0.42 (0.93) | 0.0000 | 0.34 (0.85) | 0.34 (0.89) | 0.0000 | 0.37 (0.87) | 0.37 (0.90) | 0.0000 |
| 00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.87) | 0.00 (0.90) | 0.0000 |
| 0.16 (0.53) | 0.18 (0.61) | -0.0350 | 0.78 (2.88) | 0.77 (2.89) | 0.0035 | 0.56 (2.33) | 0.56 (2.35) | 0.0000 |
| 00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (2.33) | 0.00(2.35) | 0.0000 |
| 18 (0.6%) | 20 (0.6%) | 0.0000 | 54 (0.9%) | 53 (0.9%) | 0.0000 | 072 (0.8%) | 073 (0.8%) | 0.0000 |
| 326 (10.2%) | 347 (10.9%) | -0.0022 | 721 (12.4%) | 732 (12.6%) | -0.0006 | 1,047 (11.6%) | 1,079 (12.0%) | -0.0124 |
| 0.23 (1.14) | 0.26 (1.02) | -0.0277 | 1.72 (2.75) | 1.71 (3.02) | 0.0035 | 1.19 (2.31) | 1.20 (2.50) | -0.0042 |
| 00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.0000 | 0.65 (2.31) | 0.65 (2.50) | 0.0000 |
| 0.73 (0.59) | 0.73 (0.53) | 0.0000 | 0.49 (0.53) | 0.50 (0.54) | -0.0187 | 0.58 (0.55) | 0.58 (0.54) | 0.0000 |
| 00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.0000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.35 (0.55) | 0.35 (0.54) | 0.0000 |
| 1.35 (6.46) | 1.58 (8.51) | -0.0304 | 0.78 (2.88) | 0.77 (2.89) | 0.0035 | 0.98 (4.49) | 1.06 (5.57) | -0.0158 |
| 00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (4.49) | 0.00 (5.57) | 0.0000 |
| 462 (77.00/) | 2 446 (76 50/) | 0.0006 | 2.004 (25.00/) | 2.006 (26.00/) | 0.0002 | 4 546 (50 40/) | 4 5 42 (50 40/) | 0.0000 |
| ,402 (77.0%) | 2,440 (70.5%) | 0.0006 | 2,084 (33.8%) | 2,090 (30.0%) | -0.0003 | 4,346 (30.4%) | 4,342 (30.4%) | 0.0000 |
| 0.55 (1.10) | 0.57 (1.15) | -0.0178 | 0.22 (0.71) | 0.21 (0.71) | 0.0141 | 0.34 (0.87) | 0.34 (0.89) | 0.0000 |
| 00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.87) | 0.00 (0.89) | 0.0000 |
| 205 (12 40/) | 401 (12 50/) | 0.0002 | 752 (12 00/) | 762 (12 10/) | 0.0006 | 1 147 (12 79/) | 1 164 (12 00/) | -0.0060 |
| 393 (12.4%) | 401 (12.5%) | -0.0003 | 732 (12.970) | /03 (13.170) | -0.0000 | 1,147 (12.776) | 1,104 (12.9%) | -0.0000 |
| ,172 (67.9%) | 2,175 (68.0%) | -0.0001 | 2,980 (51.2%) | 3,031 (52.1%) | -0.0013 | 5,152 (57.2%) | 5,206 (57.8%) | -0.0121 |
| 761 (23.8%) | 771 (24.1%) | -0.0006 | 1,213 (20.9%) | 1,262 (21.7%) | -0.0017 | 1,974 (21.9%) | 2,033 (22.6%) | -0.0168 |
| ,368 (42.8%) | 1,331 (41.6%) | 0.0019 | 1,458 (25.1%) | 1,429 (24.6%) | 0.0010 | 2,826 (31.4%) | 2,760 (30.6%) | 0.0173 |
| 536 (16.8%) | 505 (15.8%) | 0.0025 | 684 (11.8%) | 672 (11.6%) | 0.0006 | 1,220 (13.5%) | 1,177 (13.1%) | 0.0118 |
| 32.98 (33.52) | 32.63 (41.44) | | 21.73 (21.64) | 21.97 (23.47) | -0.0106 | 25.72 (26.47) | 25.75 (31.06) | -0.0010 |
| 0 [13.60, 40.24] | 23.21 [10.71, 40.75] | 0.0263 | 16.93 [8.43, 28.46] | 16.47 [8.00, 29.05] | 0.0204 | 19.51 (26.47) | 18.86 (31.06) | 0.0225 |
| 754 (23.6%) | 785 (24.5%) | -0.002 | N/A | N/A | N/A | 754 (23.6%) | 785 (24.5%) | -0.002 |
| ,444 (76.4%) | 2,413 (75.5%) | 0.001 | N/A | N/A | N/A | 2,444 (76.4%) | 2,413 (75.5%) | 0.001 |
| N/A | N/A | N/A | 2,179 (37.5%) | 2,153 (37.0%) | 0.001 | 2,179 (37.5%) | 2,153 (37.0%) | 0.001 |
| N/A | N/A | N/A | 636 (10.9%) | 629 (10.8%) | 0.000 | 636 (10.9%) | 629 (10.8%) | 0.000 |
| N/A | N/A | N/A | 2,686 (46.2%) | 2,711 (46.6%) | -0.001 | 2,686 (46.2%) | 2,711 (46.6%) | -0.001 |
| N/A | N/A | N/A | 315 (5.4%) | 323 (5.6%) | -0.001 | 315 (5.4%) | 323 (5.6%) | -0.001 |
| | 0.0 [6.00, 17.00]<br>0.42 (0.91)<br>0.0 [0.00, 1.00]<br>0.16 (0.53)<br>0.0 [0.00, 0.00]<br>18 (0.6%)<br>326 (10.2%)<br>0.23 (1.14)<br>00 [0.00, 0.00]<br>0.73 (0.59)<br>10 [0.00, 1.00]<br>1.35 (6.46)<br>10 [0.00, 0.00]<br>462 (77.0%)<br>0.55 (1.10)<br>10 [0.00, 1.00]<br>395 (12.4%)<br>4,172 (67.9%)<br>761 (23.8%)<br>368 (42.8%)<br>536 (16.8%)<br>1.298 (33.52)<br>0 [13.60, 40.24]<br>754 (23.6%)<br>444 (76.4%)<br>N/A<br>N/A | 00 [6.00, 17.00] 11.00 [7.00, 16.25] 0.42 (0.91) 0.42 (0.93) 00 [0.00, 1.00] 0.00 [0.00, 1.00] 0.16 (0.53) 0.18 (0.61) 00 [0.00, 0.00] 0.00 [0.00, 0.00] 18 (0.6%) 20 (0.6%) 326 (10.2%) 347 (10.9%) 0.23 (1.14) 0.26 (1.02) 00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.73 (0.59) 0.73 (0.53) 10 [0.00, 1.00] 1.58 (8.51) 00 [0.00, 0.00] 2,446 (76.5%) 0.55 (1.10) 0.57 (1.15) 00 [0.00, 1.00] 0.00 [0.00, 1.00] 395 (12.4%) 401 (12.5%) 317 (267.9%) 2,175 (68.0%) 761 (23.8%) 771 (24.1%) 3,368 (42.8%) 1,331 (41.6%) 536 (16.8%) 505 (15.8%) 22.98 (33.52) 32.63 (41.44) 0 [13.60, 40.24] 23.21 [10.71, 40.75] 754 (23.6%) 785 (24.5%) 2,443 (75.5%) N/A N/A N/A N/A N/A N/A N/A N/A N/A | 00 [6.00, 17.00] 11.00 [7.00, 16.25] -0.1087 0.42 (0.91) 0.42 (0.93) 0.0000 00 [0.00, 1.00] 0.00 [0.00, 1.00] 0.0000 0.16 (0.53) 0.18 (0.61) -0.0350 10 [0.00, 0.00] 0.00 [0.00, 0.00] 0.0000 18 (0.6%) 20 (0.6%) 0.0000 326 (10.2%) 347 (10.9%) -0.0022 0.23 (1.14) 0.26 (1.02) -0.0277 10 [0.00, 0.00] 0.00 [0.00, 0.00] 0.0000 0.73 (0.59) 0.73 (0.53) 0.0000 0.00 [0.00, 1.00] 1.00 [0.00, 1.00] 0.0000 1.35 (6.46) 1.58 (8.51) -0.0304 00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.0000 3.462 (77.0%) 2,446 (76.5%) 0.0006 0.55 (1.10) 0.57 (1.15) -0.0178 00 [0.00, 1.00] 0.00 [0.00, 1.00] 0.0000 395 (12.4%) 401 (12.5%) -0.0003 3,172 (67.9%) 2,175 (68.0%) -0.0017 761 (23.8%) 771 (24.1%) -0.006 368 (42.8%) 1,331 (41.6%) 0.0019 536 (16.8%) <td< td=""><td> 11.00 [7.00, 1.6.25]</td><td><math display="block">\begin{array}{cccccccccccccccccccccccccccccccccccc</math></td><td><math display="block">\begin{array}{c} 00 \left[ 6.00, 17.00 \right] &amp; 11.00 \left[ 7.00, 16.25 \right] &amp; -0.1087 &amp; 9.00 \left[ 5.00, 14.00 \right] &amp; 9.00 \left[ 5.00, 13.00 \right] &amp; 0.0000 \\ 0.042 \left( 0.91 \right) &amp; 0.42 \left( 0.93 \right) &amp; 0.0000 &amp; 0.34 \left( 0.85 \right) &amp; 0.34 \left( 0.89 \right) &amp; 0.0000 \\ 0.00 \left[ 0.00, 1.00 \right] &amp; 0.00 \left[ 0.00, 1.00 \right] &amp; 0.0000 &amp; 0.00 \left[ 0.00, 0.00 \right] &amp; 0.00 \left[ 0.00, 0.00 \right] &amp; 0.0000 \\ 0.016 \left( 0.53 \right) &amp; 0.18 \left( 0.61 \right) &amp; -0.0350 &amp; 0.78 \left( 2.88 \right) &amp; 0.77 \left( 2.89 \right) &amp; 0.0035 \\ 0.00 \left[ 0.00, 0.00 \right] &amp; 0.00 \left[ 0.00, 0.00 \right] &amp; 0.0000 &amp; 0.00 \left[ 0.00, 0.00 \right] &amp; 0.00 \left[ 0.00, 0.00 \right] &amp; 0.0000 \\ 18 \left( 0.6\% \right) &amp; 20 \left( 0.6\% \right) &amp; 0.0000 &amp; 34 \left( 0.9\% \right) &amp; 53 \left( 0.9\% \right) &amp; 0.0000 \\ 326 \left( 10.2\% \right) &amp; 347 \left( 10.9\% \right) &amp; -0.0022 &amp; 721 \left( 12.4\% \right) &amp; 732 \left( 12.6\% \right) &amp; -0.0006 \\ 0.023 \left( 1.14 \right) &amp; 0.26 \left( 1.02 \right) &amp; -0.0277 &amp; 1.72 \left( 2.75 \right) &amp; 1.71 \left( 3.02 \right) &amp; 0.0035 \\ 10 \left[ 0.00, 0.00 \right] &amp; 0.00 \left[ 0.00, 0.00 \right] &amp; 0.0000 &amp; 1.00 \left[ 0.00, 2.00 \right] &amp; 0.0000 \\ 0.73 \left( 0.59 \right) &amp; 0.73 \left( 0.53 \right) &amp; 0.0000 &amp; 0.49 \left( 0.53 \right) &amp; 0.50 \left( 0.54 \right) &amp; -0.0187 \\ 10 \left[ 0.00, 0.01 \right] &amp; 1.00 \left[ 0.00, 1.00 \right] &amp; 0.0000 &amp; 0.00 \left[ 0.00, 1.00 \right] &amp; 0.00 \left[ 0.00, 1.00 \right] &amp; 0.000 \\ 0.00 \left[ 0.00, 0.00 \right] &amp; 0.00 \left[ 0.00, 0.00 \right] &amp; 0.0000 &amp; 0.00 \left[ 0.00, 0.00 \right] &amp; 0.00 \left[ 0.00, 0.00 \right] &amp; 0.0000 \\ 0.462 \left( 77.0\% \right) &amp; 2.446 \left( 76.5\% \right) &amp; 0.0006 &amp; 2.084 \left( 35.8\% \right) &amp; 2.096 \left( 36.0\% \right) &amp; -0.0003 \\ 0.55 \left( 1.10 \right) &amp; 0.57 \left( 1.15 \right) &amp; -0.0178 &amp; 0.22 \left( 0.71 \right) &amp; 0.21 \left( 0.71 \right) &amp; 0.0141 \\ 00 \left[ 0.00, 1.00 \right] &amp; 0.00 \left[ 0.00, 1.00 \right] &amp; 0.0000 &amp; 0.00 \left[ 0.00, 0.00 \right] &amp; 0.00 \left[ 0.00, 0.00 \right] \\ 0.00 \left[ 0.00, 1.00 \right] &amp; 0.00 \left[ 0.00, 1.00 \right] &amp; 0.0006 &amp; 1.213 \left( 20.9\% \right) &amp; 3.031 \left( 52.1\% \right) &amp; -0.0013 \\ 356 \left( 16.8\% \right) &amp; 771 \left( 24.1\% \right) &amp; -0.0006 &amp; 1.213 \left( 20.9\% \right) &amp; 3.031 \left( 52.1\% \right) &amp; -0.0013 \\ 356 \left( 16.8\% \right) &amp; 771 \left( 24.1\% \right) &amp; -0.0006 &amp; 1.213 \left( 20.9\% \right) &amp; 1.452 \left( 21.7\% \right) &amp; -0.0107 \\ 3368 \left( 42.8\% \right) &amp; 771 \left( 24.1\% \right) &amp; -0.0006 &amp; 1.213 \left( 20.9\% \right) &amp; 1.262 \left( 21.7\% \right) &amp; -0.0017 \\ 3368 \left( 42.8\% \right) &amp; 771 \left( 24.1\% \right) &amp; -0.0006 &amp; 1.213 \left( 20.9\% \right) &amp; 1.262 \left( 21.7\% \right) &amp; -0.0017 \\ 3368 \left( 42.8\% \right) &amp; 7331 \left( 14.6\% \right) &amp; 0.0025 &amp; 684 \left( </math></td><td><math display="block">\begin{array}{c} 0[(6.00,17.00] &amp; 11.00[7.00,16.25] &amp; -0.1087 &amp; 9.00[5.00,14.00] &amp; 9.00[5.00,13.00] &amp; 0.0000 &amp; 9.35(8.24) \\ 0.42(0.91) &amp; 0.42(0.93) &amp; 0.0000 &amp; 0.34(0.85) &amp; 0.34(0.89) &amp; 0.0000 &amp; 0.37(0.87) \\ 0.10(0.00,1.00] &amp; 0.00[0.00,1.00] &amp; 0.0000 &amp; 0.00[0.00,0.00] &amp; 0.00[0.00,0.00] &amp; 0.0000 &amp; 0.00[0.87] \\ 0.16(0.53) &amp; 0.18(0.61) &amp; -0.0350 &amp; 0.78(2.88) &amp; 0.77(2.89) &amp; 0.0035 &amp; 0.56(2.33) \\ 0.16(0.63) &amp; 20(0.6%) &amp; 0.0000 &amp; 0.00[0.00,0.00] &amp; 0.00[0.00,0.00] &amp; 0.0000 &amp; 0.00(2.33) \\ 18(0.6\%) &amp; 20(0.6\%) &amp; 0.0000 &amp; 54(0.9\%) &amp; 53(0.9\%) &amp; 0.0000 &amp; 0.72(0.8\%) \\ 326(10.2\%) &amp; 347(10.9\%) &amp; -0.0022 &amp; 721(12.4\%) &amp; 732(12.6\%) &amp; -0.0006 &amp; 1.047(11.6\%) \\ 0.23(1.14) &amp; 0.26(1.02) &amp; -0.0277 &amp; 1.72(2.75) &amp; 1.71(3.02) &amp; 0.0035 &amp; 1.19(2.31) \\ 00(0.00,0.00] &amp; 0.00(0.00,0.00] &amp; 0.0000 &amp; 1.00(0.00,0.00] &amp; 1.00(0.00,0.00] &amp; 0.0000 &amp; 0.65(2.31) \\ 00(0.00,0.00] &amp; 0.07(0.59) &amp; 0.73(0.53) &amp; 0.0000 &amp; 0.49(0.53) &amp; 0.50(0.54) &amp; -0.0187 &amp; 0.58(0.55) \\ 00(0.00,1.00] &amp; 1.00(0.00,1.00] &amp; 0.0000 &amp; 0.00(0.00,1.00] &amp; 0.00(0.00,0.00] &amp; 0.0000 &amp; 0.35(0.55) \\ 1.135(6.46) &amp; 1.58(8.51) &amp; -0.0304 &amp; 0.78(2.88) &amp; 0.77(2.89) &amp; 0.0035 &amp; 0.98(4.49) \\ 00(0.00,0.00] &amp; 0.00(0.00,0.00] &amp; 0.0000 &amp; 0.00(0.00,0.00] &amp; 0.00(0.00,0.00] &amp; 0.0000 &amp; 0.34(6.65) \\ 0.55(1.10) &amp; 0.57(1.15) &amp; -0.0178 &amp; 0.22(0.71) &amp; 0.21(0.71) &amp; 0.0141 &amp; 0.34(0.87) \\ 0.00(0.00,1.00] &amp; 0.00(0.00,1.00] &amp; 0.0000 &amp; 0.00(0.00,0.00] &amp; 0.00(0.00,0.00] &amp; 0.000 &amp; 0.00(0.87) \\ 395(12.4\%) &amp; 401(12.5\%) &amp; -0.0005 &amp; 2.980(51.2\%) &amp; 3.031(52.1\%) &amp; -0.0013 &amp; 5,152(57.2\%) \\ 701(23.8\%) &amp; 771(24.1\%) &amp; -0.0006 &amp; 1.213(2.09\%) &amp; 1.262(21.7\%) &amp; -0.0013 &amp; 5,152(57.2\%) \\ 715(23.8\%) &amp; 771(24.1\%) &amp; -0.0006 &amp; 1.213(2.09\%) &amp; 1.262(21.7\%) &amp; -0.0016 &amp; 1.297(23.647) \\ 0(13.60,40.24) &amp; 2.131(41.6\%) &amp; 0.0013 &amp; 1.438(25.1\%) &amp; 1.647(20.9\%) &amp; 0.0006 &amp; 1.220(13.5\%) \\ 0(13.60,40.24) &amp; 2.413(75.5\%) &amp; 0.0025 &amp; 684(11.8\%) &amp; 672(11.6\%) &amp; 0.0001 &amp; 2.797(37.5\%) \\ 0(13.60,40.24) &amp; 2.413(75.5\%) &amp; 0.001 &amp; N/A &amp; N/A &amp; N/A &amp; N/A &amp; N/A &amp; N/A &amp; N/A &amp; N/A &amp; </math></td><td><math display="block">\begin{array}{c} 0_10(6,00,17.00) &amp; 11.00 &amp; (7.00,16.25) &amp; -0.1087 &amp; 9.00 &amp; (5.00,14.00) &amp; 9.00 &amp; (5.00,13.00) &amp; 0.0000 &amp; 9.35 &amp; (8.24) &amp; 9.71 &amp; (7.78) \\ 0.42 &amp; (0.91) &amp; 0.42 &amp; (0.93) &amp; 0.0000 &amp; 0.34 &amp; (0.85) &amp; 0.34 &amp; (0.89) &amp; 0.0000 &amp; 0.00 &amp; 0.00 &amp; (0.87) &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 &amp; 0.00 </math></td></td<> | 11.00 [7.00, 1.6.25] | $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | $\begin{array}{c} 00 \left[ 6.00, 17.00 \right] & 11.00 \left[ 7.00, 16.25 \right] & -0.1087 & 9.00 \left[ 5.00, 14.00 \right] & 9.00 \left[ 5.00, 13.00 \right] & 0.0000 \\ 0.042 \left( 0.91 \right) & 0.42 \left( 0.93 \right) & 0.0000 & 0.34 \left( 0.85 \right) & 0.34 \left( 0.89 \right) & 0.0000 \\ 0.00 \left[ 0.00, 1.00 \right] & 0.00 \left[ 0.00, 1.00 \right] & 0.0000 & 0.00 \left[ 0.00, 0.00 \right] & 0.00 \left[ 0.00, 0.00 \right] & 0.0000 \\ 0.016 \left( 0.53 \right) & 0.18 \left( 0.61 \right) & -0.0350 & 0.78 \left( 2.88 \right) & 0.77 \left( 2.89 \right) & 0.0035 \\ 0.00 \left[ 0.00, 0.00 \right] & 0.00 \left[ 0.00, 0.00 \right] & 0.0000 & 0.00 \left[ 0.00, 0.00 \right] & 0.00 \left[ 0.00, 0.00 \right] & 0.0000 \\ 18 \left( 0.6\% \right) & 20 \left( 0.6\% \right) & 0.0000 & 34 \left( 0.9\% \right) & 53 \left( 0.9\% \right) & 0.0000 \\ 326 \left( 10.2\% \right) & 347 \left( 10.9\% \right) & -0.0022 & 721 \left( 12.4\% \right) & 732 \left( 12.6\% \right) & -0.0006 \\ 0.023 \left( 1.14 \right) & 0.26 \left( 1.02 \right) & -0.0277 & 1.72 \left( 2.75 \right) & 1.71 \left( 3.02 \right) & 0.0035 \\ 10 \left[ 0.00, 0.00 \right] & 0.00 \left[ 0.00, 0.00 \right] & 0.0000 & 1.00 \left[ 0.00, 2.00 \right] & 0.0000 \\ 0.73 \left( 0.59 \right) & 0.73 \left( 0.53 \right) & 0.0000 & 0.49 \left( 0.53 \right) & 0.50 \left( 0.54 \right) & -0.0187 \\ 10 \left[ 0.00, 0.01 \right] & 1.00 \left[ 0.00, 1.00 \right] & 0.0000 & 0.00 \left[ 0.00, 1.00 \right] & 0.00 \left[ 0.00, 1.00 \right] & 0.000 \\ 0.00 \left[ 0.00, 0.00 \right] & 0.00 \left[ 0.00, 0.00 \right] & 0.0000 & 0.00 \left[ 0.00, 0.00 \right] & 0.00 \left[ 0.00, 0.00 \right] & 0.0000 \\ 0.462 \left( 77.0\% \right) & 2.446 \left( 76.5\% \right) & 0.0006 & 2.084 \left( 35.8\% \right) & 2.096 \left( 36.0\% \right) & -0.0003 \\ 0.55 \left( 1.10 \right) & 0.57 \left( 1.15 \right) & -0.0178 & 0.22 \left( 0.71 \right) & 0.21 \left( 0.71 \right) & 0.0141 \\ 00 \left[ 0.00, 1.00 \right] & 0.00 \left[ 0.00, 1.00 \right] & 0.0000 & 0.00 \left[ 0.00, 0.00 \right] & 0.00 \left[ 0.00, 0.00 \right] \\ 0.00 \left[ 0.00, 1.00 \right] & 0.00 \left[ 0.00, 1.00 \right] & 0.0006 & 1.213 \left( 20.9\% \right) & 3.031 \left( 52.1\% \right) & -0.0013 \\ 356 \left( 16.8\% \right) & 771 \left( 24.1\% \right) & -0.0006 & 1.213 \left( 20.9\% \right) & 3.031 \left( 52.1\% \right) & -0.0013 \\ 356 \left( 16.8\% \right) & 771 \left( 24.1\% \right) & -0.0006 & 1.213 \left( 20.9\% \right) & 1.452 \left( 21.7\% \right) & -0.0107 \\ 3368 \left( 42.8\% \right) & 771 \left( 24.1\% \right) & -0.0006 & 1.213 \left( 20.9\% \right) & 1.262 \left( 21.7\% \right) & -0.0017 \\ 3368 \left( 42.8\% \right) & 771 \left( 24.1\% \right) & -0.0006 & 1.213 \left( 20.9\% \right) & 1.262 \left( 21.7\% \right) & -0.0017 \\ 3368 \left( 42.8\% \right) & 7331 \left( 14.6\% \right) & 0.0025 & 684 \left( $ | $\begin{array}{c} 0[(6.00,17.00] & 11.00[7.00,16.25] & -0.1087 & 9.00[5.00,14.00] & 9.00[5.00,13.00] & 0.0000 & 9.35(8.24) \\ 0.42(0.91) & 0.42(0.93) & 0.0000 & 0.34(0.85) & 0.34(0.89) & 0.0000 & 0.37(0.87) \\ 0.10(0.00,1.00] & 0.00[0.00,1.00] & 0.0000 & 0.00[0.00,0.00] & 0.00[0.00,0.00] & 0.0000 & 0.00[0.87] \\ 0.16(0.53) & 0.18(0.61) & -0.0350 & 0.78(2.88) & 0.77(2.89) & 0.0035 & 0.56(2.33) \\ 0.16(0.63) & 20(0.6%) & 0.0000 & 0.00[0.00,0.00] & 0.00[0.00,0.00] & 0.0000 & 0.00(2.33) \\ 18(0.6\%) & 20(0.6\%) & 0.0000 & 54(0.9\%) & 53(0.9\%) & 0.0000 & 0.72(0.8\%) \\ 326(10.2\%) & 347(10.9\%) & -0.0022 & 721(12.4\%) & 732(12.6\%) & -0.0006 & 1.047(11.6\%) \\ 0.23(1.14) & 0.26(1.02) & -0.0277 & 1.72(2.75) & 1.71(3.02) & 0.0035 & 1.19(2.31) \\ 00(0.00,0.00] & 0.00(0.00,0.00] & 0.0000 & 1.00(0.00,0.00] & 1.00(0.00,0.00] & 0.0000 & 0.65(2.31) \\ 00(0.00,0.00] & 0.07(0.59) & 0.73(0.53) & 0.0000 & 0.49(0.53) & 0.50(0.54) & -0.0187 & 0.58(0.55) \\ 00(0.00,1.00] & 1.00(0.00,1.00] & 0.0000 & 0.00(0.00,1.00] & 0.00(0.00,0.00] & 0.0000 & 0.35(0.55) \\ 1.135(6.46) & 1.58(8.51) & -0.0304 & 0.78(2.88) & 0.77(2.89) & 0.0035 & 0.98(4.49) \\ 00(0.00,0.00] & 0.00(0.00,0.00] & 0.0000 & 0.00(0.00,0.00] & 0.00(0.00,0.00] & 0.0000 & 0.34(6.65) \\ 0.55(1.10) & 0.57(1.15) & -0.0178 & 0.22(0.71) & 0.21(0.71) & 0.0141 & 0.34(0.87) \\ 0.00(0.00,1.00] & 0.00(0.00,1.00] & 0.0000 & 0.00(0.00,0.00] & 0.00(0.00,0.00] & 0.000 & 0.00(0.87) \\ 395(12.4\%) & 401(12.5\%) & -0.0005 & 2.980(51.2\%) & 3.031(52.1\%) & -0.0013 & 5,152(57.2\%) \\ 701(23.8\%) & 771(24.1\%) & -0.0006 & 1.213(2.09\%) & 1.262(21.7\%) & -0.0013 & 5,152(57.2\%) \\ 715(23.8\%) & 771(24.1\%) & -0.0006 & 1.213(2.09\%) & 1.262(21.7\%) & -0.0016 & 1.297(23.647) \\ 0(13.60,40.24) & 2.131(41.6\%) & 0.0013 & 1.438(25.1\%) & 1.647(20.9\%) & 0.0006 & 1.220(13.5\%) \\ 0(13.60,40.24) & 2.413(75.5\%) & 0.0025 & 684(11.8\%) & 672(11.6\%) & 0.0001 & 2.797(37.5\%) \\ 0(13.60,40.24) & 2.413(75.5\%) & 0.001 & N/A & $ | $\begin{array}{c} 0_10(6,00,17.00) & 11.00 & (7.00,16.25) & -0.1087 & 9.00 & (5.00,14.00) & 9.00 & (5.00,13.00) & 0.0000 & 9.35 & (8.24) & 9.71 & (7.78) \\ 0.42 & (0.91) & 0.42 & (0.93) & 0.0000 & 0.34 & (0.85) & 0.34 & (0.89) & 0.0000 & 0.00 & 0.00 & (0.87) & 0.00 $ |

<sup>\*</sup>Included in the 1:1 PS matching model

Optum (PS matched): https://bwh-dope.aetion.com/projects/details/1406/results/63149/result/44 Marketscan (PS matched): https://bwh-dope.aetion.com/projects/details/1407/results/63153/result/44